CLINICAL TRIAL: NCT00379769
Title: A Long Term, Open Label, Randomised Study in Patients With Type 2 Diabetes, Comparing the Combination of Rosiglitazone and Either Metformin or Sulfonylurea With Metformin Plus Sulfonylurea on Cardiovascular Endpoints and Glycaemia
Brief Title: RECORD: Rosiglitazone Evaluated for Cardiac Outcomes and Regulation of Glycaemia in Diabetes
Acronym: RECORD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRL-049653/231
Record Dates: First submitted 2006-09-21; First posted 2006-09-22 (Estimated); Results first posted 2009-11-13 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; CV outcomes; rosiglitazone; Type II diabetes; sulfonylurea; RECORD; metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Rosiglitazone; Sulfonylurea Compounds; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- rosiglitazone in addition to background metformin (Experimental): Participants inadequately controlled on background metformin (MET) were randomised to receive rosiglitazone (RSG), in addition to MET. RSG was initiated as a 4 mg once daily dose and was increased to a maximum dose of 8 mg per day as required to achieve a target HbA1c of less than or equal to 7.0 percent.
  Interventions: Drug: Rosiglitazone; Drug: Metformin
- rosiglitazone in addition to background sulfonylurea (Experimental): Participants inadequately controlled on background SU were randomised to receive, in addition to SU, RSG. RSG was initiated as a 4 mg once daily dose and was increased to a maximum dose of 8 mg per day as required to achieve a target HbA1c of less than or equal to 7.0 percent.
  Interventions: Drug: Rosiglitazone; Drug: Sulfonylurea
- Sulfonylurea in addition to background metformin (Active Comparator): Participants inadequately controlled on background MET were randomised to receive, in addition to MET, a sulfonylurea (SU) (glibenclamide, gliclazide, or glimepiride). The SU was gradually increased to the maximum permitted dose (glibenclamide 15 mg per day or miconizied equivalent of 10.5 mg per day; gliclazide 240 mg per day; glimepiride 4 mg per day) as required to achieve a target HbA1c of less than or equal to 7.0 percent.
  Interventions: Drug: Sulfonylurea; Drug: Metformin
- Metformin in addition to background sulfonylurea (Active Comparator): Participants inadequately controlled on background SU were randomised to receive, in addition to SU, MET. MET was gradually increased to the maximum permitted dose of 2550 mg per day as required to achieve a target HbA1c of less than or equal to 7.0 percent.
  Interventions: Drug: Sulfonylurea; Drug: Metformin

INTERVENTIONS:
Drug: Rosiglitazone — Rosiglitazone maximum 8 mg per day
  Arms: rosiglitazone in addition to background metformin; rosiglitazone in addition to background sulfonylurea
Drug: Sulfonylurea — Sulfonylurea (SU) maximum permitted daily dose
  Arms: Metformin in addition to background sulfonylurea; Sulfonylurea in addition to background metformin; rosiglitazone in addition to background sulfonylurea
Drug: Metformin — Metformin maximum permitted daily dose .
  Arms: Metformin in addition to background sulfonylurea; Sulfonylurea in addition to background metformin; rosiglitazone in addition to background metformin

SUMMARY:
This study is a phase 3b, multicentre, randomised, open label, parallel group study. A 4-week run-in period will be followed by a median of 6 years of treatment with study medication in addition to continuation of background glucose lowering therapy. Patients inadequately controlled on background metformin will be randomised to receive, in addition to metformin, either rosiglitazone or a sulfonylurea(glibenclamide, gliclazide or glimepiride) in a ratio of 1:1. Patients inadequately controlled on background SU will be randomised to receive, in addition to SU, either rosiglitazone or metformin in a ratio of 1:1. Equal numbers of patients receiving background metformin and SU at entry will be entered into the study.

DETAILED DESCRIPTION:
A RECORD follow-up study is being performed to monitor the incidence of cancer and bone fractures in RECORD patients for a period of 4 years after the end of the main RECORD study (2008 - 2012).

ELIGIBILITY:
Inclusion Criteria:

* Patients with type II diabetes mellitus as defined by 1999 World Health Organisation criteria.
* Glycated haemoglobin (HbA1c) >7.0 % to = 9.0 % at visit 1.
* Use of an oral glucose lowering agent for a minimum of 6 months prior to screening and unchanged for 2 months prior to screening.
* Body mass index >25.0 kg/m2.

Exclusion Criteria:

* Patients receiving any other glucose lowering therapy which is not metformin or a sulfonylurea.
* Patients with systolic blood pressure >180 mmHg or diastolic blood pressure >105 mmHg.
* Patients who have required the use of insulin for glycaemic control at any time in the past.
* Hospitalisation for any major cardiovascular event in the last 3 months.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4447 (Actual)
Dates: Start 2001-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (373):
- Australia (11):
  - GSK Investigational Site, Miranda, New South Wales
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Wollongong, New South Wales
  - GSK Investigational Site, Carina Heights, Queensland
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Sherwood, Queensland
  - GSK Investigational Site, Keswick, South Australia
  - GSK Investigational Site, North Adelaide, South Australia
  - GSK Investigational Site, Port Lincoln, South Australia
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Malvern, Victoria
- Belgium (13):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Arlon
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Genk
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Kortrijk
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Moerkerke
  - GSK Investigational Site, Oostham
  - GSK Investigational Site, Roeselare
  - GSK Investigational Site, Sint-Gillis-Waas
  - GSK Investigational Site, Vilvoorde
- Bulgaria (4):
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- Croatia (5):
  - GSK Investigational Site, Krapinske Toplice
  - GSK Investigational Site, Rijeka
  - GSK Investigational Site, Slavonski Brod
  - GSK Investigational Site, Varaždin
  - GSK Investigational Site, Zagreb
- Czechia (11):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, České Budějovice
  - GSK Investigational Site, Holice V Cechach
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Jindřichův Hradec
  - GSK Investigational Site, Ostrava Poruba
  - GSK Investigational Site, Písek
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Rakovník
  - GSK Investigational Site, Tábor
  - GSK Investigational Site, Trutnov
- Denmark (12):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Aarhus
  - GSK Investigational Site, Copenhagen
  - GSK Investigational Site, Glostrup Municipality
  - GSK Investigational Site, Hilleroed
  - GSK Investigational Site, Kolding
  - GSK Investigational Site, København NV
  - GSK Investigational Site, Køge
  - GSK Investigational Site, Næstved
  - GSK Investigational Site, Odense C
  - GSK Investigational Site, Silkeborg
  - GSK Investigational Site, Slagelse
- Estonia (7):
  - GSK Investigational Site, Paide
  - GSK Investigational Site, Pärnu
  - GSK Investigational Site, Rakvere
  - GSK Investigational Site, Saku
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
  - GSK Investigational Site, Viljandi
- Finland (15):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Hanko
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Hyvinkää
  - GSK Investigational Site, Jyväskylä
  - GSK Investigational Site, Kerava
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Lahti
  - GSK Investigational Site, Lappeenranta
  - GSK Investigational Site, Oulun Kaupunki
  - GSK Investigational Site, Riihimäki
  - GSK Investigational Site, Rovaniemi
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- France (75):
  - GSK Investigational Site, Bully-les-Mines, Hauts-de-France
  - GSK Investigational Site, Amilly
  - GSK Investigational Site, Arras
  - GSK Investigational Site, Aspach-le-Bas
  - GSK Investigational Site, Aubagne
  - GSK Investigational Site, Auchy-lès-Hesdin
  - GSK Investigational Site, Azille
  - GSK Investigational Site, Beaumont-le-Roger
  - GSK Investigational Site, Beaumont-sur-Lèze
  - GSK Investigational Site, Belfort
  - GSK Investigational Site, Belpech
  - GSK Investigational Site, Blotzheim
  - GSK Investigational Site, Bondy
  - GSK Investigational Site, BP 1542 Dijon
  - GSK Investigational Site, Broglie
  - GSK Investigational Site, Calmont
  - GSK Investigational Site, Carbonne
  - GSK Investigational Site, Carcassonne
  - GSK Investigational Site, Cassis
  - GSK Investigational Site, Castelnaudary
  - GSK Investigational Site, Catelnaudary
  - GSK Investigational Site, Cernay
  - GSK Investigational Site, Champhol
  - GSK Investigational Site, Chartres
  - GSK Investigational Site, Colmar
  - GSK Investigational Site, Corbeil Essonne
  - GSK Investigational Site, Coursan
  - GSK Investigational Site, Cuincy
  - GSK Investigational Site, Danjoutin
  - GSK Investigational Site, Dessenheim
  - GSK Investigational Site, Dieppe
  - GSK Investigational Site, Dunkirk
  - GSK Investigational Site, Épernon
  - GSK Investigational Site, Gémenos
  - GSK Investigational Site, Hanches
  - GSK Investigational Site, Hautot-sur-Mer
  - GSK Investigational Site, Husseren-Wesserling
  - GSK Investigational Site, Kembs
  - GSK Investigational Site, La Barre-en-Ouche
  - GSK Investigational Site, La Verdière
  - GSK Investigational Site, Labarth-Sur-Leze
  - GSK Investigational Site, Labarthe-sur-Lèze
  - GSK Investigational Site, Le Grau-du-Roi
  - GSK Investigational Site, Le Lherm 31600
  - GSK Investigational Site, Le Perray-en-Yvelines
  - GSK Investigational Site, Lezignan-Corbières
  - GSK Investigational Site, Maintenon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Masevaux
  - GSK Investigational Site, Maubeuge
  - GSK Investigational Site, Monfort Sur Risle
  - GSK Investigational Site, Mulhouse
  - GSK Investigational Site, Muret
  - GSK Investigational Site, Nassandres
  - GSK Investigational Site, Nevers
  - GSK Investigational Site, Nogent-le-Phaye
  - GSK Investigational Site, Orbec
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pierre-Bénite
  - GSK Investigational Site, Pierres
  - GSK Investigational Site, Pinsaguel
  - GSK Investigational Site, Roux Mesnil Bouteille
  - GSK Investigational Site, Rugles
  - GSK Investigational Site, Saint Leger Sur Yvelines
  - GSK Investigational Site, Saint-Eulalie Badens
  - GSK Investigational Site, Seysses
  - GSK Investigational Site, Thann
  - GSK Investigational Site, Thiberville
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Trebbes
  - GSK Investigational Site, Trèbes
  - GSK Investigational Site, Valenciennes
  - GSK Investigational Site, Vogelsheim
  - GSK Investigational Site, Voves
  - GSK Investigational Site, Wittenheim
- Germany (24):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Sinsheim, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Kronach, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Kronberg, Hesse
  - GSK Investigational Site, Ober-Mörlen, Hesse
  - GSK Investigational Site, Offenbach, Hesse
  - GSK Investigational Site, Wetzlar, Hesse
  - GSK Investigational Site, Bad Lauterberg im Harz, Lower Saxony
  - GSK Investigational Site, Beckum, North Rhine-Westphalia
  - GSK Investigational Site, Menden, North Rhine-Westphalia
  - GSK Investigational Site, Gau-Algesheim, Rhineland-Palatinate
  - GSK Investigational Site, Kallstadt, Rhineland-Palatinate
  - GSK Investigational Site, Lambrecht, Rhineland-Palatinate
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Speyer, Rhineland-Palatinate
  - GSK Investigational Site, Friedrichsthal, Saarland
  - GSK Investigational Site, Burgstädt, Saxony
  - GSK Investigational Site, Chemnitz, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Suhl, Thuringia
- Greece (8):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Haidari, Athens
  - GSK Investigational Site, Ioannina
  - GSK Investigational Site, Marousi
  - GSK Investigational Site, Pátrai
  - GSK Investigational Site, Piraeus-Athens
  - GSK Investigational Site, Thessaloniki
  - GSK Investigational Site, Thessalonikis
- Hungary (13):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Eger
  - GSK Investigational Site, Győr
  - GSK Investigational Site, Gyula
  - GSK Investigational Site, Kurtag99
  - GSK Investigational Site, Nyiregyháza
  - GSK Investigational Site, Patkaj98
  - GSK Investigational Site, Siófok
  - GSK Investigational Site, Szentes
  - GSK Investigational Site, Szombathely
  - GSK Investigational Site, Veszprém
  - GSK Investigational Site, Zalaegerszeg
- Italy (21):
  - GSK Investigational Site, Reggio Calabria, Calabria
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Nocera Inferiore (SA), Campania
  - GSK Investigational Site, Salerno, Campania
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Rimini, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Brescia, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, San Donato (MI), Lombardy
  - GSK Investigational Site, Treviglio (BG), Lombardy
  - GSK Investigational Site, Campobasso, Molise
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Cagliari, Sardinia
  - GSK Investigational Site, Sassari, Sardinia
  - GSK Investigational Site, Palermo, Sicily
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Bari
  - GSK Investigational Site, Parma
  - GSK Investigational Site, Roma
- Latvia (7):
  - GSK Investigational Site, Jēkabpils
  - GSK Investigational Site, Lagzdi60
  - GSK Investigational Site, Limbaži
  - GSK Investigational Site, Ogre
  - GSK Investigational Site, Riga
  - GSK Investigational Site, Sturii59
  - GSK Investigational Site, Tukums
- Lithuania (3):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Klaipėda
  - GSK Investigational Site, Vilnius
- Netherlands (16):
  - GSK Investigational Site, Geleen
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Hengelo
  - GSK Investigational Site, Hoogvliet
  - GSK Investigational Site, Kerkrade
  - GSK Investigational Site, Landgraaf
  - GSK Investigational Site, Musselkanaal
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Oude Pekela
  - GSK Investigational Site, Ridderkerk
  - GSK Investigational Site, Rijswijk
  - GSK Investigational Site, Roosendaal
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Sint Willebrord
  - GSK Investigational Site, Zoetermeer
  - GSK Investigational Site, Zwijndrecht
- New Zealand (8):
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Dunedin
  - GSK Investigational Site, Hastings
  - GSK Investigational Site, Otahuhu, Auckland
  - GSK Investigational Site, Palmerston North
  - GSK Investigational Site, Takapuna, Auckland
  - GSK Investigational Site, Tauranga
  - GSK Investigational Site, Wellington
- Poland (11):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Grudziądz
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Romania (5):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Timișoara
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- Slovakia (12):
  - GSK Investigational Site, Banská Bystrica
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Košice
  - GSK Investigational Site, Kysucké Nové Mesto
  - GSK Investigational Site, Lučenec
  - GSK Investigational Site, Ľubochňa
  - GSK Investigational Site, Prešov
  - GSK Investigational Site, Prievidza
  - GSK Investigational Site, Šahy
  - GSK Investigational Site, Šamorín
  - GSK Investigational Site, Trenčín
  - GSK Investigational Site, Žilina
- Spain (13):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Benidorm
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Cadiz
  - GSK Investigational Site, Cáceres
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Reus
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Vazquc56
  - GSK Investigational Site, Vizcaya
- Sweden (19):
  - GSK Investigational Site, Eksjö
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Helsingborg
  - GSK Investigational Site, Köping
  - GSK Investigational Site, Kristianstad
  - GSK Investigational Site, Kungälv
  - GSK Investigational Site, Linköpiing
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Mora
  - GSK Investigational Site, Nacka
  - GSK Investigational Site, Norrköping
  - GSK Investigational Site, Oskarshamn
  - GSK Investigational Site, Skene
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uddevalla
  - GSK Investigational Site, Umeå
  - GSK Investigational Site, Uppsala
  - GSK Investigational Site, Vadstena
- Ukraine (6):
  - GSK Investigational Site, Dnipro
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lviv
  - GSK Investigational Site, Vinnitsa
- United Kingdom (52):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Fowley, Cornwall
  - GSK Investigational Site, Chesterfield, Derbyshire
  - GSK Investigational Site, Airdrie, Lanarkshire
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Hamilton, Lanarkshire
  - GSK Investigational Site, Motherwell, Lanarkshire
  - GSK Investigational Site, Leicester, Leicestershire
  - GSK Investigational Site, Northampton, Northamptonshire
  - GSK Investigational Site, Linwood, Renfrewshire
  - GSK Investigational Site, Paisley, Renfrewshire
  - GSK Investigational Site, Frome, Somerset
  - GSK Investigational Site, Glastonbury, Somerset
  - GSK Investigational Site, Rugby, Warwickshire
  - GSK Investigational Site, Corsham, Wiltshire
  - GSK Investigational Site, Trowbridge, Wiltshire
  - GSK Investigational Site, Westbury, Wiltshire
  - GSK Investigational Site, Airdrie
  - GSK Investigational Site, Ashford
  - GSK Investigational Site, Bath
  - GSK Investigational Site, Chesterfield
  - GSK Investigational Site, Chippenham
  - GSK Investigational Site, Coatbridge
  - GSK Investigational Site, Colney
  - GSK Investigational Site, Cumbernauld
  - GSK Investigational Site, Dronfield
  - GSK Investigational Site, Dumbarton
  - GSK Investigational Site, East Kilbride
  - GSK Investigational Site, Falmouth
  - GSK Investigational Site, Garston, Watford
  - GSK Investigational Site, Gateshead
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Hamilton
  - GSK Investigational Site, Harrow
  - GSK Investigational Site, Kirkintilloch
  - GSK Investigational Site, Leigh-on-Sea
  - GSK Investigational Site, Motherwell
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Newport
  - GSK Investigational Site, Nottingham
  - GSK Investigational Site, Old Whittington, Chesterfield
  - GSK Investigational Site, Paisley
  - GSK Investigational Site, Penzance
  - GSK Investigational Site, Rubery, Birmingham
  - GSK Investigational Site, Sheffield
  - GSK Investigational Site, Thornhill
  - GSK Investigational Site, Thornhill, Cardiff
  - GSK Investigational Site, Uddingston
  - GSK Investigational Site, Weston-super-Mare
  - GSK Investigational Site, Wishaw
  - GSK Investigational Site, Woking
  - GSK Investigational Site, Worle, Weston-Super-Mare

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Home PD, Jones NP, Pocock SJ, Beck-Nielsen H, Gomis R, Hanefeld M, Komajda M, Curtis P; RECORD Study Group. Rosiglitazone RECORD study: glucose control outcomes at 18 months. Diabet Med. 2007 Jun;24(6):626-34. doi: 10.1111/j.1464-5491.2007.02160.x. PMID 17517066
- [Background] Home PD, Pocock SJ, Beck-Nielsen H, Gomis R, Hanefeld M, Dargie H, Komajda M, Gubb J, Biswas N, Jones NP. Rosiglitazone Evaluated for Cardiac Outcomes and Regulation of Glycaemia in Diabetes (RECORD): study design and protocol. Diabetologia. 2005 Sep;48(9):1726-35. doi: 10.1007/s00125-005-1869-1. Epub 2005 Jul 16. PMID 16025252
- [Background] Home PD, Pocock SJ, Beck-Nielsen H, Gomis R, Hanefeld M, Jones NP, Komajda M, McMurray JJ; RECORD Study Group. Rosiglitazone evaluated for cardiovascular outcomes--an interim analysis. N Engl J Med. 2007 Jul 5;357(1):28-38. doi: 10.1056/NEJMoa073394. Epub 2007 Jun 5. PMID 17551159
- [Background] Home PD, Pocock SJ, Beck-Nielsen H, Curtis PS, Gomis R, Hanefeld M, Jones NP, Komajda M, McMurray JJ; RECORD Study Team. Rosiglitazone evaluated for cardiovascular outcomes in oral agent combination therapy for type 2 diabetes (RECORD): a multicentre, randomised, open-label trial. Lancet. 2009 Jun 20;373(9681):2125-35. doi: 10.1016/S0140-6736(09)60953-3. Epub 2009 Jun 6. PMID 19501900
- [Background] Komajda M, Curtis P, Hanefeld M, Beck-Nielsen H, Pocock SJ, Zambanini A, Jones NP, Gomis R, Home PD; RECORD Study Group. Effect of the addition of rosiglitazone to metformin or sulfonylureas versus metformin/sulfonylurea combination therapy on ambulatory blood pressure in people with type 2 diabetes: a randomized controlled trial (the RECORD study). Cardiovasc Diabetol. 2008 Apr 24;7:10. doi: 10.1186/1475-2840-7-10. PMID 18435852
- [Derived] Jones NP, Curtis PS, Home PD. Cancer and bone fractures in observational follow-up of the RECORD study. Acta Diabetol. 2015 Jun;52(3):539-46. doi: 10.1007/s00592-014-0691-y. Epub 2014 Dec 19. PMID 25524432
- [Derived] MacDonald MR, Petrie MC, Home PD, Komajda M, Jones NP, Beck-Nielsen H, Gomis R, Hanefeld M, Pocock SJ, Curtis PS, McMurray JJ. Incidence and prevalence of unrecognized myocardial infarction in people with diabetes: a substudy of the Rosiglitazone Evaluated for Cardiac Outcomes and Regulation of Glycemia in Diabetes (RECORD) study. Diabetes Care. 2011 Jun;34(6):1394-6. doi: 10.2337/dc10-2398. Epub 2011 May 11. PMID 21562320
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: BRL-049653/231 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: BRL-049653/231 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: BRL-049653/231 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: BRL-049653/231 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: BRL-049653/231 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: BRL-049653/231 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: BRL-049653/231 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The RECORD study ran from April 2001 through December 2008. Results are presented in the non-re-adjudicated outcome measures (OMs). An independent patient-level re-adjudication of mortality, non-fatal myocardial infarction, and non-fatal stroke began on January 2011 and ran through March 2012. The results are presented in the re-adjudicated OMs.
Pre-assignment Details: The RECORD observational follow-up (OFU) started at the end of the RECORD study and ran through December 2012. OFU was designed to collect cancer and bone fracture data. Participants were not provided with study medication in the OFU. Data are presented for the entire study (RECORD + OBF) and for OFU alone in the observational OMs.
Groups:
- RSG in Addition to Background MET: Participants inadequately controlled on background metformin (MET) were randomised to receive rosiglitazone (RSG), in addition to MET. RSG was initiated as a 4 mg once daily dose and was increased to a maximum dose of 8 mg per day as required to achieve a target HbA1c of less than or equal to 7.0 percent.
- SU in Addition to Background MET: Participants inadequately controlled on background MET were randomised to receive, in addition to MET, a sulfonylurea (SU) (glibenclamide, gliclazide, or glimepiride). The SU was gradually increased to the maximum permitted dose (glibenclamide 15 mg per day or micronized equivalent of 10.5 mg per day; gliclazide 240 mg per day; glimepiride 4 mg per day) as required to achieve a target HbA1c of less than or equal to 7.0 percent.
- RSG in Addition to Background SU: Participants inadequately controlled on background SU were randomised to receive, in addition to SU, RSG. RSG was initiated as a 4 mg once daily dose and was increased to a maximum dose of 8 mg per day as required to achieve a target HbA1c of less than or equal to 7.0 percent.
- MET in Addition to Background SU: Participants inadequately controlled on background SU were randomised to receive, in addition to SU, MET. MET was gradually increased to the maximum permitted dose of 2550 mg per day as required to achieve a target HbA1c of less than or equal to 7.0 percent.
- Combined RSG: Observational Follow-up: Participants randomized to receive RSG (MET+RSG and SU+RSG) in the main RECORD study. Participants were not provided with study medication in the observational follow-up; instead, anti-diabetic treatment was prescribed at the investigator's discretion.
- Combined MET/SU: Observational Follow-up: Participants randomized to the active control groups (MET+SU and SU+MET) in the main RECORD study. Participants were not provided with study medication in the observational follow-up; instead, anti-diabetic treatment was prescribed at the investigator's discretion.
Period: Main Study
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU | Combined RSG: Observational Follow-up | Combined MET/SU: Observational Follow-up
Started | 1117 | 1105 | 1103 | 1122 | 0 | 0
Completed | 939 | 906 | 896 | 892 | 0 | 0
Not Completed | 178 | 199 | 207 | 230 | 0 | 0
Not completed — Death | 57 | 67 | 54 | 72 | 0 | 0
Not completed — Adverse Event | 5 | 8 | 10 | 11 | 0 | 0
Not completed — Lost to Follow-up | 29 | 29 | 25 | 26 | 0 | 0
Not completed — Withdrawal by Subject | 46 | 56 | 72 | 70 | 0 | 0
Not completed — Moved to survival status follow-up only | 27 | 25 | 32 | 36 | 0 | 0
Not completed — Participant moved | 3 | 2 | 3 | 3 | 0 | 0
Not completed — Poor compliance | 3 | 2 | 2 | 1 | 0 | 0
Not completed — Prohibited glucose lowering medication | 0 | 3 | 0 | 1 | 0 | 0
Not completed — Site closed | 4 | 4 | 4 | 8 | 0 | 0
Not completed — Entry criteria violation | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Participant did not take study drug | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 2 | 1 | 1 | 0 | 0
Not completed — Participant completed study at visit 27 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Personal reasons | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Risk of heart failure | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Investigator refused to log temperature | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Reason unspecified | 0 | 0 | 1 | 0 | 0 | 0
Period: Observational Follow-up
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU | Combined RSG: Observational Follow-up | Combined MET/SU: Observational Follow-up
Started | 0 | 0 | 0 | 0 | 1280 (665 from "RSG in Addition to Background MET" arm; 615 from "RGS in Addition to Background SU" arm.) | 1250 (647 from "SU in Addition to Background MET" arm; 603 from "MET in Addition to Background SU" arm.)
Completed | 0 | 0 | 0 | 0 | 1131 | 1102
Not Completed | 0 | 0 | 0 | 0 | 149 | 148
Not completed — Death | 0 | 0 | 0 | 0 | 78 | 70
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 25 | 27
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 12 | 12
Not completed — Entered into Another Clinical Trial | 0 | 0 | 0 | 0 | 18 | 22
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 8 | 8
Not completed — Site Closed Early | 0 | 0 | 0 | 0 | 6 | 7
Not completed — Participant Moved | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Unknown; Reason Not Provided | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU | Total
Number analyzed (Participants) | 1117 | 1105 | 1103 | 1122 | 4447
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (8.02) | 57.2 (8.14) | 59.8 (8.26) | 59.7 (8.23) | 58.4 (8.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 516 | 521 | 562 | 554 | 2153
  Male | 601 | 584 | 541 | 568 | 2294
Race/Ethnicity, Customized [Number; unit: participants]
  White | 1105 | 1087 | 1095 | 1112 | 4399
  Black | 3 | 6 | 2 | 3 | 14
  Oriental | 4 | 2 | 5 | 7 | 18
  Aboriginal | 1 | 0 | 0 | 0 | 1
  African | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 2 | 1 | 0 | 4
  Egyptian | 1 | 0 | 0 | 0 | 1
  Gipsy | 1 | 0 | 0 | 0 | 1
  Indian | 0 | 1 | 0 | 0 | 1
  Maori | 0 | 1 | 0 | 0 | 1
  Middle East Hible | 0 | 1 | 0 | 0 | 1
  Pacific Islander | 0 | 1 | 0 | 0 | 1
  Polynesian | 0 | 1 | 0 | 0 | 1
  Sri Lankan | 0 | 2 | 0 | 0 | 2
  Tahitian | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cardiovascular Death/Cardiovascular Hospitalisation Events
Description: The number of participants with cardiovascular death events (death due to cardiovascular causes or deaths with insufficient information to rule out a cardiovascular cause) and cardiovascular hospitalisation events (hospitalisation for a cardiovascular event, excluding planned admissions not associated with a worsening of the disease/condition of the participant) was recorded.
Time Frame: Baseline through End of Study (up to 7.5 years)
Population: Intent-to-Treat (ITT) Population: all randomized participants who were treated with at least one dose of study medication
Measure: Number; unit: participants
Groups:
- Combined RSG: Participants inadequately controlled on background MET or background SU were randomised to receive RSG, in addition to MET or SU. RSG was initiated as a 4 mg once daily dose and was increased to a maximum dose of 8 mg per day as required to achieve a target HbA1c of less than or equal to 7.0 percent.
- Combined MET/SU: Participants inadequately controlled on background MET were randomised to receive, in addition to MET, an SU (glibenclamide, gliclazide, or glimepiride). The SU was gradually increased to the maximum permitted dose (glibenclamide 15 mg per day or micronized equivalent of 10.5 mg per day; gliclazide 240 mg per day; glimepiride 4 mg per day) as required to achieve a target HbA1c of less than or equal to 7.0 percent. Participants inadequately controlled on background SU were randomised to receive, in addition to SU, MET. MET was gradually increased to the maximum permitted dose of 2550 mg per day as required to achieve a target HbA1c of less than or equal to 7.0 percent.
Arm/Group | Combined RSG | Combined MET/SU
Number analyzed (Participants) | 2220 | 2227
participants | 321 | 323
Statistical Analysis 1: Comparison: Combined RSG vs Combined MET/SU; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of 1.2 for the upper limit of the 95 percent confidence interval in time to event analysis comparing RSG to MET/SU stratified by background medication; Hazard Ratio (HR) = 0.99, 95% CI [0.85 to 1.16]

2. Secondary Outcome: Number of Participants With Cardiovascular Events and All-cause Deaths
Description: Composites of participants with first cardiovascular (CV) hospitalisations and CV death or all-cause death and individual first events of acute myocardial infarction (MI) , stroke, congestive heart failure (CHF), CV death, and all-cause death.
Time Frame: Baseline through End of Study (up to 7.5 years)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Combined RSG | Combined MET/SU
Number analyzed (Participants) | 2220 | 2227
participants
  CV death, acute MI, stroke | 154 | 165
  CV death, acute MI, stroke, unstable angina | 171 | 184
  CV death, acute MI, stroke, unstable angina, CHF | 204 | 206
  All-cause death,acuteMI,stroke,unstable angina,CHF | 251 | 268
  Acute MI (fatal or non-fatal) | 64 | 56
  Stroke (fatal or non-fatal) | 46 | 63
  CHF (fatal or non-fatal) | 61 | 29
  Death from CV causes | 60 | 71
  Death (all cause) during CV follow-up | 111 | 139
  Death (all-cause) including survival status | 136 | 157

3. Secondary Outcome: Total Number of Cardiovascular Hospitalisations and Cardiovascular Deaths
Description: The total number of events for individual components of cardiovascular (CV) hospitalisations and cardiovascular deaths were recorded. MI, myocardial infarction.
Time Frame: Baseline through End of Study (up to 7.5 years)
Population: as for outcome 1
Measure: Number; unit: Number of events
Arm/Group | Combined RSG | Combined MET/SU
Number analyzed (Participants) | 2220 | 2227
Number of events
  CV deaths | 60 | 71
  Death due to acute MI | 7 | 10
  Death due to heart failure | 10 | 2
  Sudden death | 8 | 12
  Death due to acute vascular events | 1 | 10
  Other CV mortality | 6 | 4
  Death of presumed CV cause | 28 | 33
  Cardiovascular hospitalisation | 483 | 490
  Hospitalisation for acute MI | 66 | 57
  Hospitalisation for unstable angina | 28 | 28
  Hospitalisation for congestive heart failure | 69 | 36
  Hospitalisation for stroke | 51 | 67
  Hospitalisation for transient ischaemic attack | 10 | 10
  Hospitalisation for invasive CV procedure | 99 | 116
  Hospitalisation for amputation of extremities | 6 | 23
  Other CV hospitalisations | 154 | 153

4. Secondary Outcome: Number of Participants With First Cardiovascular Hospitalisations/Cardiovascular Deaths by Stratum
Description: Participants with first cardiovascular death (death due to cardiovascular causes or deaths with insufficient information to rule out a cardiovascular cause) and cardiovascular hospitalisation (hospitalisation for a cardiovascular event, excluding planned admissions not associated with a worsening of the disease/condition of the participant) were recorded by study stratum.
Time Frame: Baseline through End of Study (up to 7.5 years)
Population: as for outcome 1
Measure: Number; unit: partcipants
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU
Number analyzed (Participants) | 1117 | 1105 | 1103 | 1122
partcipants | 158 | 154 | 163 | 169

5. Secondary Outcome: Number of Participants With CV/Microvascular Events
Description: The number of participants with first cardiovascular or microvascular events (renal, foot, eye) were recorded.
Time Frame: Baseline through End of Study (up to 7.5 years)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Combined RSG | Combined MET/SU
Number analyzed (Participants) | 2220 | 2227
participants
  Participants with a CV/Microvascular event | 363 | 385
  Participants with any microvascular event | 59 | 78
  Participants with any eye event | 42 | 52
  Participants with any foot event | 19 | 28
  Participants with any renal event | 0 | 0

6. Secondary Outcome: Number of Participants With Glycaemic Failure Events
Description: Failure of glycaemic control was defined as two consecutive HbA1c values of ≥8.5 percent, or HbA1c ≥8.5percent at a single visit, after which the subject was either moved to the post-randomised treatment phase or triple therapy was started.
Time Frame: Baseline through to end of randomised dual therapy
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU
Number analyzed (Participants) | 1117 | 1105 | 1103 | 1122
participants | 281 | 451 | 365 | 424

7. Secondary Outcome: Number of Participants With Addition of Third Oral Agent/Switch to Insulin
Description: The number of participants with addition of a third oral agent or switch to insulin from randomised dual combination treatment were recorded.
Time Frame: Baseline through End of Study (up to 7.5 years)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU
Number analyzed (Participants) | 1117 | 1105 | 1103 | 1122
participants
  Participants with an event | 295 | 183 | 344 | 171
  First Event - Triple Therapy | 257 | 7 | 296 | 6
  First Event - Insulin | 38 | 176 | 49 | 165

8. Secondary Outcome: The Number of Participants Starting Insulin at Any Time During the Study
Description: The number of participants starting insulin at any time during the study was recorded.
Time Frame: Baseline through End of Study (up to 7.5 years)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU
Number analyzed (Participants) | 1117 | 1105 | 1103 | 1122
participants | 126 | 276 | 168 | 259

9. Secondary Outcome: Model Adjusted Change From Baseline in HbA1c at Month 60
Description: Model adjusted (adjusted for any imbalances in the baseline values between within stratum treatment groups) change from baseline in HbA1c was calculated as the value at Month 60 minus the Baseline value.
Time Frame: Baseline and Month 60 of randomised dual therapy treatment period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU
Number analyzed (Participants) | 1096 | 1079 | 1073 | 1079
Percent | -0.14 (0.035) | 0.17 (0.042) | -0.24 (0.039) | -0.10 (0.039)

10. Secondary Outcome: Model Adjusted Change From Baseline in Fasting Plasma Glucose at Month 60
Description: Model adjusted (adjusted for any imbalances in the baseline values between within stratum treatment groups) change from baseline in fasting plasma glucose was calculated as the value at Month 60 minus the Baseline value.
Time Frame: Baseline to Month 60 of the randomised dual therapy treatment period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmol/L (millimoles/Liter)
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU
Number analyzed (Participants) | 1095 | 1078 | 1074 | 1079
mmol/L (millimoles/Liter) | -1.38 (0.073) | -0.29 (0.090) | -2.00 (0.085) | -0.94 (0.094)

11. Secondary Outcome: Model Adjusted Mean Change From Baseline in Insulin and Pro-insulin at Month 60
Description: Model adjusted (adjusted for any imbalances in the baseline values between within stratum treatment groups) change from baseline in insulin and pro-insulin was calculated as the value at Month 60 minus the Baseline value.
Time Frame: Baseline to Month 60 of the randomised dual therapy treatment period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: picamoles/liter (pmol/L)
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU
Number analyzed (Participants) | 931 | 982 | 882 | 940
picamoles/liter (pmol/L)
  Insulin, Adjusted Change from Baseline | -18.6 (1.01) | 3.7 (1.77) | -16.9 (1.65) | -12.1 (1.91)
  Pro-insulin, Adjusted Change from Baseline | -2.4 (0.26) | 4.2 (0.43) | -3.2 (0.48) | -3.0 (0.37)

12. Secondary Outcome: Number of HbA1c and Fasting Plasma Glucose (FPG) Responders at Month 60
Description: Number of responders, i.e., participants meeting glycaemic targets (HbA1c less than or equal to 7 percent, FPG less than or equal to 7 mmol/L)
Time Frame: Baseline to Month 60 of the randomised dual therapy treatment period
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU
Number analyzed (Participants) | 1117 | 1105 | 1103 | 1122
participants
  HbA1c Responders | 265 | 208 | 235 | 180
  FPG Responders | 300 | 180 | 257 | 154

13. Secondary Outcome: Model Adjusted Ratio to Baseline (Expressed as a Percentage) Homeostasis Model Assessment (HOMA) Beta Cell Function and Insulin Sensitivity at Month 60
Description: The model adjusted (adjusted for any imbalances in the baseline [BL] values between within stratum treatment groups) ratio to BL in HOMA beta-cell function and insulin sensitivity was calculated as the ratio of the Month 60 value to the BL value and was expressed as percent change from BL. For each treatment group, the model-adjusted mean change from BL at Month 60 was determined on the log scale. This mean was then back transformed to give a geometric mean (GM) of the ratio of the Month 60 value to BL on the original scale. The GM was expressed as a percentage (100*[GM^-1]).
Time Frame: Baseline to Month 60 of the randomised dual therapy treatment phase
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU
Number analyzed (Participants) | 926 | 977 | 878 | 933
percent change
  Beta cell function | 20.54 [16.52 to 24.70] | 19.28 [14.66 to 24.09] | 32.35 [26.55 to 38.41] | 12.43 [7.42 to 17.67]
  Insulin sensitivity | 42.57 [37.57 to 47.76] | -3.45 [-7.21 to 0.47] | 42.07 [36.39 to 47.98] | 23.90 [19.36 to 28.61]

14. Secondary Outcome: Model Adjusted Ratio to Baseline (Expressed as a Percentage) for Total Cholesterol (TC), Low-density Lipoprotein (LDL) Cholesterol, High-density Lipoprotein (HDL) Cholesterol, Triglycerides, and Free Fatty Acids (FFAs) at Month 60
Description: The model adjusted (adjusted for any imbalances in the baseline [BL] values between within stratum treatment groups) ratio to BL in TC, LDL cholesterol, HDL cholesterol, triglycerides, and FFAs was calculated as the ratio of the Month 60 value to the BL value and was expressed as percent change from BL. For each treatment group, the model-adjusted mean change from BL at Month 60 was determined on the log scale. This mean was then back transformed to give a geometric mean (GM) of the ratio of the Month 60 value to BL on the original scale. The GM was expressed as a percentage (100*[GM^-1]).
Time Frame: Baseline to Month 60 of the randomised dual therapy treatment phase
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU
Number analyzed (Participants) | 1117 | 1105 | 1103 | 1122
percent change
  Total cholesterol | -5.49 [-6.99 to -3.96] | -9.09 [-10.33 to -7.84] | -2.91 [-4.62 to -1.17] | -9.68 [-11.03 to -8.31]
  HDL-cholesterol | 9.95 [8.44 to 11.49] | 2.57 [1.46 to 3.68] | 7.73 [6.18 to 9.30] | 6.14 [4.88 to 7.42]
  LDL-cholesterol | -12.70 [-15.03 to -10.30] | -17.68 [-19.70 to -15.61] | -8.99 [-11.42 to -6.49] | -17.80 [-19.93 to -15.61]
  Triglycerides | -7.97 [-10.72 to -5.15] | -1.95 [-4.73 to 0.91] | -2.68 [-5.69 to 0.43] | -2.50 [-5.21 to 0.28]
  Free fatty acids | -16.46 [-19.13 to -13.71] | 2.79 [-0.23 to 5.91] | -11.58 [-14.65 to -8.41] | 4.47 [1.23 to 7.81]

15. Secondary Outcome: Model Adjusted Ratio to Baseline (Expressed as a Percentage) for Total Cholesterol (TC):High-density Lipoprotein (HDL) Cholesterol and Low-density Lipoprotein (LDL) Cholesterol:HDL Cholesterol Ratios at Month 60
Description: The model adjusted (adjusted for any imbalances in the baseline [BL] values between within stratum treatment groups) ratio to BL in TC:HDL cholesterol and LDL cholesterol:HDL cholesterol was calculated as the ratio of the Month 60 value to the BL value and was expressed as percent change from BL. For each treatment group, the model-adjusted mean change from BL at Month 60 was determined on the log scale. This mean was then back transformed to give a geometric mean (GM) of the ratio of the Month 60 value to BL on the original scale. The GM was expressed as a percentage (100*[GM^-1]).
Time Frame: Baseline to Month 60 of the randomised dual therapy treatment period
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU
Number analyzed (Participants) | 1117 | 1105 | 1103 | 1122
percent change
  Total Cholesterol: HDL Cholesterol Ratio | -14.20 [-15.98 to -12.39] | -11.33 [-12.82 to -9.81] | -9.93 [-11.83 to -7.98] | -15.01 [-16.44 to -13.55]
  LDL Cholesterol: HDL-Cholesterol Ratio | -20.89 [-23.24 to -18.46] | -20.04 [-22.16 to -17.87] | -15.85 [-18.26 to -13.37] | -22.53 [-24.63 to -20.37]

16. Secondary Outcome: Model Adjusted Ratio to Baseline (Expressed as a Percentage) for Apolipoprotein B (Apo-B) at Month 60
Description: The model adjusted (adjusted for any imbalances in the baseline [BL] values between within stratum treatment groups) ratio to BL in Apo-B was calculated as the ratio of the Month 60 value to the BL value and was expressed as percent change from BL. For each treatment group, the model-adjusted mean change from BL at Month 60 was determined on the log scale. This mean was then back transformed to give a geometric mean (GM) of the ratio of the Month 60 value to BL on the original scale. The GM was expressed as a percentage (100*[GM^-1]).
Time Frame: Baseline to Month 60 of the randomised dual therapy treatment period
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU
Number analyzed (Participants) | 949 | 1007 | 906 | 970
percent change | -13.77 [-15.45 to -12.05] | -11.63 [-13.10 to -10.14] | -9.68 [-11.55 to -7.77] | -12.09 [-13.67 to -10.47]

17. Secondary Outcome: Model Adjusted Ratio to Baseline (Expressed as a Percentage) for Urinary Albumin Creatinine Ratio at Month 60
Description: The model adjusted (adjusted for any imbalances in the baseline [BL] values between within stratum treatment groups) ratio to BL in urinary albumin creatinine ratio was calculated as the ratio of the Month 60 value to the BL value and was expressed as percent change from BL. For each treatment group, the model-adjusted mean change from BL at Month 60 was determined on the log scale. This mean was then back transformed to give a geometric mean (GM) of the ratio of the Month 60 value to BL on the original scale. The GM was expressed as a percentage (100*[GM^-1]).
Time Frame: Baseline to Month 60 of the randomised dual therapy treatment phase
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU
Number analyzed (Participants) | 899 | 921 | 891 | 901
percent change | 8.31 [-0.70 to 18.14] | 15.17 [6.73 to 24.28] | -3.43 [-11.91 to 5.87] | 11.91 [3.10 to 21.46]

18. Secondary Outcome: Model Adjusted Change From Baseline in Body Weight at Month 60
Description: Model adjusted (adjusted for any imbalances in the baseline values between within stratum treatment groups) change from baseline in body weight was calculated as the value at Month 60 minus the Baseline value.
Time Frame: Baseline to Month 60 of the randomised dual therapy treatment phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: kilograms
Groups:
- RSG in Addition to Background MET: Participants inadequately controlled on background MET were randomised to receive RSG, in addition to MET. RSG was initiated as a 4 mg once daily dose and was increased to a maximum dose of 8 mg per day as required to achieve a target HbA1c of less than or equal to 7.0 percent.
- SU in Addition to Background MET: Participants inadequately controlled on background MET were randomised to receive, in addition to MET, an SU (glibenclamide, gliclazide, or glimepiride). The SU was gradually increased to the maximum permitted dose (glibenclamide 15 mg per day or miconizied equivalent of 10.5 mg per day; gliclazide 240 mg per day; glimepiride 4 mg per day) as required to achieve a target HbA1c of less than or equal to 7.0 percent.
- RSG in Addition to Background SU: Participants inadequately controlled on background SU were randomised to receive, in addition to SU, RSG. RSG was initiated as a 4 mg once daily dose and was increased to a maximum dose of 8mg per day as required to achieve a target HbA1c of less than or equal to 7.0 percent.
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU
Number analyzed (Participants) | 1096 | 1079 | 1073 | 1079
kilograms | 3.93 (0.263) | -0.54 (0.192) | 4.72 (0.235) | -2.16 (0.179)

19. Secondary Outcome: Model Adjusted Change From Baseline in Alanine Aminotransferase at Month 60
Description: Model adjusted (adjusted for any imbalances in the baseline values between within stratum treatment groups) change from baseline in alanine aminotransferase was calculated as the value at Month 60 minus the Baseline value.
Time Frame: Baseline to Month 60 of the randomised dual therapy treatment phase
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: U/L (Units/Liter)
Groups:
- SU in Addition to Background MET: Participants inadequately controlled on background MET were randomised to receive, in addition to MET, an SU (glibenclamide, gliclazide or glimepiride). The SU was gradually increased to the maximum permitted dose (glibenclamide 15 mg per day or miconizied equivalent of 10.5 mg per day; gliclazide 240 mg per day; glimepiride 4 mg per day) as required to achieve a target HbA1c of less than or equal to 7.0 percent.
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU
Number analyzed (Participants) | 1094 | 1077 | 1073 | 1078
U/L (Units/Liter) | -37.43 [-39.22 to -35.59] | -21.73 [-23.90 to -19.50] | -30.17 [-31.98 to -28.31] | -24.00 [-26.21 to -21.73]

20. Secondary Outcome: Model Adjusted Change From Baseline in Waist Circumference at Month 60
Description: Model adjusted (adjusted for any imbalances in the baseline values between within stratum treatment groups) change from baseline in waist circumference was calculated as the value at Month 60 minus the Baseline value.
Time Frame: Baseline to Month 60 of the randomised dual therapy treatment phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: cm (centimeters)
Groups:
- RSG in Addition to Background MET: Participants inadequately controlled on background MET were randomised to receive RSG, in addition to MET. RSG was initiated as a 4mg once daily dose and was increased to a maximum dose of 8mg per day as required to achieve a target HbA1c of less than or equal to 7.0 percent.
- SU in Addition to Background MET: Participants inadequately controlled on background MET were randomised to receive, in addition to MET, an SU (glibenclamide, gliclazide or glimepiride). The SU was gradually increased to the maximum permitted dose (glibenclamide 15mg per day or miconizied equivalent of 10.5mg per day; gliclazide 240mg per day and glimepiride 4mg per day) as required to achieve a target HbA1c of less than or equal to 7.0 percent.
- RSG in Addition to Background SU: Participants inadequately controlled on background SU were randomised to receive, in addition to SU, RSG. RSG was initiated as a 4mg once daily dose and was increased to a maximum dose of 8mg per day as required to achieve a target HbA1c of less than or equal to 7.0 percent.
- MET in Addition to Background SU: Participants inadequately controlled on background SU were randomised to receive, in addition to SU, MET. MET was gradually increased to the maximum permitted dose of 2550mg per day as required to achieve a target HbA1c of less than or equal to 7.0 percent.
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU
Number analyzed (Participants) | 972 | 1032 | 926 | 994
cm (centimeters) | 2.70 (0.266) | 0.65 (0.214) | 3.00 (0.263) | -0.60 (0.215)

21. Secondary Outcome: Model Adjusted Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Month 60
Description: Model adjusted (adjusted for any imbalances in the baseline values between within treatment groups) change from baseline in SBP and DBP was calculated as the value at Month 60 minus the Baseline value.
Time Frame: Baseline to Month 60 of the randomised dual therapy treatment phase
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg (millimeters of mercury)
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU
Number analyzed (Participants) | 1096 | 1079 | 1074 | 1079
mmHg (millimeters of mercury)
  SBP | -1.9 (0.54) | -2.2 (0.52) | -2.3 (0.52) | -0.6 (0.53)
  DBP | -3.6 (0.34) | -3.4 (0.29) | -3.6 (0.31) | -2.3 (0.31)

22. Secondary Outcome: Model Adjusted Ratio to Baseline (Expressed as a Percentage) for C-Reactive Protein at Month 60
Description: The model adjusted (adjusted for any imbalances in the baseline [BL] values between within stratum treatment groups) ratio to BL in C-Reactive Protein was calculated as the ratio of the Month 60 value to the BL value and was expressed as percent change from BL. For each treatment group, the model-adjusted mean change from BL at Month 60 was determined on the log scale. This mean was then back transformed to give a geometric mean (GM) of the ratio of the Month 60 value to BL on the original scale. The GM was expressed as a percentage (100*[GM^-1]).
Time Frame: Baseline to Month 60 of the randomised dual therapy treatment phase
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU
Number analyzed (Participants) | 942 | 987 | 887 | 952
percent change | -57.40 [-60.41 to -54.15] | -28.92 [-33.71 to -23.79] | -56.50 [-61.56 to -55.21] | -36.29 [-41.03 to -31.17]

23. Secondary Outcome: Model Adjusted Ratio to Baseline (Expressed as a Percentage) for Fibrinogen at Month 60
Description: The model adjusted (adjusted for any imbalances in the baseline [BL] values between within stratum treatment groups) ratio to BL in fibrinogen was calculated as the ratio of the Month 60 value to the BL value and was expressed as percent change from BL. For each treatment group, the model-adjusted mean change from BL at Month 60 was determined on the log scale. This mean was then back transformed to give a geometric mean (GM) of the ratio of the Month 60 value to BL on the original scale. The GM was expressed as a percentage (100*[GM^-1]).
Time Frame: Baseline to Month 60 of the randomised dual therapy treatment phase
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU
Number analyzed (Participants) | 918 | 987 | 875 | 941
percent change | 2.12 [0.54 to 3.72] | 5.74 [4.22 to 7.28] | -0.23 [-1.79 to 1.35] | 3.14 [1.38 to 4.93]

24. Secondary Outcome: Model Adjusted Ratio to Baseline (Expressed as a Percentage) for Plasminogen Activator Inhibitor-1 (PAI-1) Antigen at Month 60
Description: The model adjusted (adjusted for any imbalances in the baseline [BL] values between within stratum treatment groups) ratio to BL in plasminogen activator inhibitor-1 (PAI-1) antigen was calculated as the ratio of the Month 60 value to the BL value and was expressed as percent change from BL. For each treatment group, the model-adjusted mean change from BL at Month 60 was determined on the log scale. This mean was then back transformed to give a geometric mean (GM) of the ratio of the Month 60 value to BL on the original scale. The GM was expressed as a percentage (100*[GM^-1]).
Time Frame: Baseline to Month 60 of the randomised dual therapy treatment phase
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU
Number analyzed (Participants) | 931 | 991 | 882 | 939
percent change | -9.85 [-14.42 to -5.02] | 15.01 [9.77 to 20.50] | -7.79 [-12.61 to -2.71] | -0.64 [-5.82 to 4.83]

25. Primary Outcome: Independent Re-adjudication Outcome: Number of Participants Who Died Due to Any Cause
Description: All deaths identified during the original record study and discovered after the re-adjudication efforts began were included.
Time Frame: Baseline through End of Study (up to 7.5 years)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Combined RSG | Combined MET/SU
Number analyzed (Participants) | 2220 | 2227
participants | 139 | 160
Statistical Analysis 1: Comparison: Combined RSG vs Combined MET/SU; Test type: Superiority or Other; Hazard Ratio (HR) = 0.86, 95% CI [0.68 to 1.08]

26. Primary Outcome: Independent Re-adjudication (IR) Outcome: Number of Participants With a First Occurrence of a Major Adverse Cardiovascular Event (MACE) Defined as CV (or Unknown) Death, Non-fatal MI, and Non-fatal Stroke Based on Original RECORD Endpoint Definitions
Description: IR was based on original RECORD endpoint definitions. CV death= no unequivocal non-CV cause (sudden death, death from acute vascular events, heart failure, acute MI, other CV causes, and deaths adjudicated as unknown cause). MI event=hospitalization + elevation of specific cardiac biomarkers above the upper limit of normal + cardiac ischemia symptoms/new pathological electrocardiogram findings. Stroke event=hospitalization + rapidly developed clinical signs of focal/global disturbance of cerebral function for more than 24 hours, with no apparent cause other than a vascular origin.
Time Frame: Baseline through End of Study (up to 7.5 years)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Combined RSG | Combined MET/SU
Number analyzed (Participants) | 2220 | 2227
participants | 181 | 188
Statistical Analysis 1: Comparison: Combined RSG vs Combined MET/SU; Test type: Superiority or Other; Hazard Ratio (HR) = 0.95, 95% CI [0.78 to 1.17]

27. Primary Outcome: Independent Re-adjudication Outcome: Number of Participants With a First Occurrence of a Major Adverse Cardiovascular Event (MACE) Defined as CV (or Unknown) Death, Non-fatal MI, and Non-fatal Stroke Based on Contemporary Endpoint Definitions
Description: Independent re-adjudication was based on the Standard Data Collection for Cardiovascular Trials Initiative (draft October 2011) endpoint definitions. CV death included death resulting from an acute MI; sudden cardiac death and death due to heart failure, stroke, and to other CV causes. Deaths of unknown cause were counted as CV deaths. MI was defined as evidence of myocardial necrosis in a clinical setting consistent with myocardial ischemia. Stroke was defined as an acute episode of neurological dysfunction caused by focal or global brain, spinal cord, or retinal vascular injury.
Time Frame: Baseline through End of Study (up to 7.5 years)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Combined RSG | Combined MET/SU
Number analyzed (Participants) | 2220 | 2227
participants | 186 | 191
Statistical Analysis 1: Comparison: Combined RSG vs Combined MET/SU; Test type: Superiority or Other; Hazard Ratio (HR) = 0.97, 95% CI [0.79 to 1.18]

28. Primary Outcome: Independent Re-adjudication Outcome: Number of Participants With a CV (or Unknown) Death, Based on Original RECORD Endpoint Definitions
Description: The number of participants with a CV death (or unknown) as determined by independent re-adjudication using the original RECORD endpoint definitions was recorded. CV death was defined as any death for which an unequivocal non-CV cause could not be established. CV death included death following heart failure, death following acute myocardial infarction (MI), sudden death, death due to acute vascular events, and other CV causes. Deaths due to unknown causes were classified as "unknown deaths," but were counted as CV deaths for the analysis of this endpoint.
Time Frame: Baseline through End of Study (up to 7.5 years)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Combined RSG | Combined MET/SU
Number analyzed (Participants) | 2220 | 2227
participants | 88 | 96
Statistical Analysis 1: Comparison: Combined RSG vs Combined MET/SU; Test type: Superiority or Other; Hazard Ratio (HR) = 0.90, 95% CI [0.68 to 1.21]

29. Primary Outcome: Independent Re-adjudication Outcome: Number of Participants With a CV (or Unknown) Death, Based on Contemporary Endpoint Definitions
Description: The number of participants with a CV (or unknown) death as determined by independent re-adjudication using the Standard Data Collection for Cardiovascular Trials Initiative (draft October 2011) endpoint definitions was recorded. CV death included death resulting from an acute myocardial infarction (MI), sudden cardiac death, death due to heart failure, death due to stroke, and death due to other CV causes. Deaths of unknown cause were counted as CV deaths.
Time Frame: Baseline through End of Study (up to 7.5 years)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Combined RSG | Combined MET/SU
Number analyzed (Participants) | 2220 | 2227
participants | 88 | 96
Statistical Analysis 1: Comparison: Combined RSG vs Combined MET/SU; Test type: Superiority or Other; Hazard Ratio (HR) = 0.90, 95% CI [0.68 to 1.21]

30. Primary Outcome: Independent Re-adjudication Outcome: Number of Participants With an Event of Myocardial Infarction (Fatal and Non-fatal), Based on Original RECORD Endpoint Definitions
Description: The number of participants with an MI (fatal or non-fatal) event as determined by independent re-adjudication using the original RECORD endpoint definitions was recorded. An event of MI was defined as hospitalization plus elevation of cardiac biomarkers troponin (TN) I and/or TNT above the upper limit of normal (ULN) or creatinine kinase (CK) MB (M=muscle type; B=brain type) isoenzyme >= 2x the ULN or CK > 2x the ULN plus typical symptoms of cardiac ischemia or new pathological electrocardiogram findings, or cause of death adjudicated as MI.
Time Frame: Baseline through End of Study (up to 7.5 years)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Combined RSG | Combined MET/SU
Number analyzed (Participants) | 2220 | 2227
participants | 68 | 60
Statistical Analysis 1: Comparison: Combined RSG vs Combined MET/SU; Test type: Superiority or Other; Hazard Ratio (HR) = 1.13, 95% CI [0.80 to 1.59]

31. Primary Outcome: Independent Re-adjudication Outcome: Number of Participants With an Event of Myocardial Infarction (Fatal and Non-fatal), Based on Contemporary Endpoint Definitions
Description: The number of participants with an MI (fatal or non-fatal) event as determined by independent re-adjudication using the Standard Data Collection for Cardiovascular Trials Initiative (draft October 2011) endpoint definitions was recorded. An event of MI was defined as evidence of myocardial necrosis in a clinical setting consistent with myocardial ischemia.
Time Frame: Baseline through End of Study (up to 7.5 years)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Combined RSG | Combined MET/SU
Number analyzed (Participants) | 2220 | 2227
participants | 72 | 62
Statistical Analysis 1: Comparison: Combined RSG vs Combined MET/SU; Test type: Superiority or Other; Hazard Ratio (HR) = 1.15, 95% CI [0.82 to 1.62]

32. Primary Outcome: Independent Re-adjudication Outcome: Number of Participants (Par.) With an Event of Stroke (Fatal and Non-fatal), Based on Original RECORD Endpoint Definitions
Description: Par. with a stroke (fatal or non-fatal) event as determined by independent re-adjudication using the original RECORD endpoint definitions was recorded. A stroke event=hospitalization plus rapidly developed clinical signs of focal (or global) disturbance of cerebral function lasting more than 24 hours (unless interrupted by thrombolysis, surgery, or death), with no apparent cause other than a vascular origin, including par. presenting clinical signs/symptoms suggestive of subarachnoid haemorrhage/intracerebral haemorrhage/cerebral ischemic necrosis or cause of death adjudicated as stroke.
Time Frame: Baseline through End of Study (up to 7.5 years)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Combined RSG | Combined MET/SU
Number analyzed (Participants) | 2220 | 2227
participants | 50 | 63
Statistical Analysis 1: Comparison: Combined RSG vs Combined MET/SU; Test type: Superiority or Other; Hazard Ratio (HR) = 0.79, 95% CI [0.54 to 1.14]

33. Primary Outcome: Independent Re-adjudication Outcome: Number of Participants With an Event of Stroke (Fatal and Non-fatal), Based on Contemporary Endpoint Definitions
Description: The number of participants with a stroke (fatal or non-fatal) event as determined by independent re-adjudication using the Standard Data Collection for Cardiovascular Trials Initiative (draft October 2011) endpoint definitions was recorded. An event of stroke was defined as an acute episode of neurological dysfunction caused by focal or global brain, spinal cord, or retinal vascular injury.
Time Frame: Baseline through End of Study (up to 7.5 years)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Combined RSG | Combined MET/SU
Number analyzed (Participants) | 2220 | 2227
participants | 53 | 64
Statistical Analysis 1: Comparison: Combined RSG vs Combined MET/SU; Test type: Superiority or Other; Hazard Ratio (HR) = 0.82, 95% CI [0.57 to 1.18]

34. Secondary Outcome: Number of Participants With the Indicated Type of Neoplasm/Cancer Event Reported as a Serious Adverse Event (SAE) or Death: Main Study + Observational Follow-up Combined
Description: The observational follow-up was designed to collect data concerning cancer and bone fractures in RECORD participants during a 4-year period after the end of the main RECORD study. At the end of the main study, all study medication was stopped. Participants were not provided with study medication in the observational follow-up; instead, anti-diabetic treatment was prescribed at the investigator's discretion. An SAE is defined as any event that is fatal; life threatening; disabling/incapacitating; results in hospitalization (excluding elective surgery or routine clinical procedures); prolongs a hospital stay; is associated with a congenital abnormality; cancer; is associated with an overdose. In addition, any event that the investigator regards as serious or that would suggest any significant hazard, contraindication, side effect, or precaution that may be associated with the study procedures should be reported as an SAE.
Time Frame: From the beginning of the main study through the end of the observational follow-up (up to 11.4 years)
Population: ITT Population. Analyses were performed by the original randomized treatment in the main RECORD study (referred to as Combined RSG and Combined MET/SU).
Measure: Number; unit: participants
Groups:
- Combined RSG: Main Study and Observational Follow-up: Participants randomized to receive RSG (MET+RSG and SU+RSG) in the main RECORD study. Participants were not provided with study medication in the observational follow-up; instead, anti-diabetic treatment was prescribed at the investigator's discretion.
- Combined MET/SU: Main Study and Observational Follow-up: Participants randomized to the active control groups (MET+SU and SU+MET) in the main RECORD study. Participants were not provided with study medication in the observational follow-up; instead, anti-diabetic treatment was prescribed at the investigator's discretion.
Arm/Group | Combined RSG: Main Study and Observational Follow-up | Combined MET/SU: Main Study and Observational Follow-up
Number analyzed (Participants) | 2220 | 2227
participants
  All neoplasms/cancer (N/C) (benign/malignant) | 196 | 215
  Malignant (Mal.) N/C | 179 | 195
  Mal. N/C; excluding non-melanomatous skin cancers | 164 | 186

35. Secondary Outcome: Number of Participants With the Indicated Type of Neoplasm/Cancer Event Reported as a Serious Adverse Event (SAE) or Death: Observational Follow-up
Description: as for outcome 34
Time Frame: From the end of the RECORD study through the end of the observational follow-up (up to 4.0 years)
Population: Observational Follow-up Population: all participants from the ITT Population of the RECORD study who provided data during the observational follow-up. Analyses were performed by the original randomized treatment in the main RECORD study (referred to as Combined RSG and Combined MET/SU).
Measure: Number; unit: participants
Arm/Group | Combined RSG: Observational Follow-up | Combined MET/SU: Observational Follow-up
Number analyzed (Participants) | 1280 | 1250
participants
  All neoplasms/cancer (N/C) (benign/malignant) | 60 | 51
  Malignant (Mal.) N/C | 59 | 51
  Mal. N/C; excluding non-melanomatous skin cancers | 55 | 46

36. Secondary Outcome: Number of Participants With the Indicated Type of Malignant Neoplasms/Cancer Events Reported as an SAE or Death by Location (Including Location of Special Interest): Main Study + Observational Follow-up Combined
Description: The observational follow-up (OFU) was designed to collect data concerning cancer and bone fractures in RECORD participants during a 4-year period after the end of the main RECORD study. At the end of the main study, all study medication was stopped. Participants were not provided with study medication in the OFU. The neoplasms/cancer events of bladder, breast, colon, liver, pancreatic, prostate cancer, and melanoma were pre-specified as cancers of interest for the OFU. An SAE is defined as any event that is fatal; life threatening; disabling/incapacitating; results in hospitalization (excluding elective surgery or routine clinical procedures); prolongs a hospital stay; is associated with a congenital abnormality; cancer; is associated with an overdose. In addition, any event that the investigator regards as serious or that would suggest any significant hazard, contraindication, side effect, or precaution that may be associated with the study procedures should be reported as an SAE.
Time Frame: From the beginning of the main study through the end of the observational follow-up (up to 11.4 years)
Population: as for outcome 34
Measure: Number; unit: participants
Arm/Group | Combined RSG: Main Study and Observational Follow-up | Combined MET/SU: Main Study and Observational Follow-up
Number analyzed (Participants) | 2220 | 2227
participants
  Any genitourinary | 57 | 57
  Prostate | 22 | 22
  Renal | 12 | 9
  Uterine | 11 | 16
  Bladder | 8 | 5
  Vaginal/vulvar | 1 | 1
  Ovarian | 5 | 4
  Any gastrointestinal | 48 | 62
  Colon/rectal cancer | 22 | 30
  Colon | 14 | 21
  Gastric | 13 | 5
  Pancreatic | 5 | 16
  Liver | 4 | 5
  Gall bladder/biliary | 4 | 5
  Gastrointestinal; not specified | 0 | 1
  Any hematologic | 12 | 6
  Lung | 19 | 15
  Skin (non-melanomatous) | 19 | 13
  Skin (melanomatous) | 6 | 4
  Metastases | 12 | 18
  Breast | 12 | 23
  Head and neck | 4 | 7
  Neurologic | 3 | 3
  Endocrine | 3 | 6
  Not specified | 0 | 1
  Other | 0 | 3

37. Secondary Outcome: Number of Participants With the Indicated Type of Malignant Neoplasms/Cancer Events Reported as an SAE or Death by Location (Including Location of Special Interest): Observational Follow-up
Description: as for outcome 36
Time Frame: From the end of the RECORD study through the end of the observational follow-up (up to 4.0 years)
Population: as for outcome 35
Measure: Number; unit: participants
Arm/Group | Combined RSG: Observational Follow-up | Combined MET/SU: Observational Follow-up
Number analyzed (Participants) | 1280 | 1250
participants
  Any genitourinary | 18 | 8
  Prostate | 7 | 1
  Renal | 5 | 2
  Uterine | 4 | 4
  Bladder | 2 | 0
  Vaginal/vulvar | 0 | 1
  Ovarian | 0 | 0
  Any gastrointestinal | 17 | 19
  Colon/rectal cancer | 5 | 11
  Colon | 2 | 7
  Gastric | 5 | 1
  Pancreatic | 4 | 3
  Liver | 2 | 2
  Gall bladder/biliary | 1 | 1
  Gastrointestinal; not specified | 0 | 1
  Any hematologic | 6 | 1
  Lung | 6 | 6
  Skin (non-melanomatous) | 6 | 5
  Skin (melanomatous) | 3 | 2
  Metastases | 3 | 6
  Breast | 2 | 7
  Head and neck | 2 | 1
  Neurologic | 1 | 1
  Endocrine | 0 | 1
  Not specified | 0 | 0
  Other | 0 | 0

38. Secondary Outcome: Number of Participants Who Died Due to the Indicated Cancer-related Event: Main Study + Observational Follow-up Combined
Description: as for outcome 34
Time Frame: From the beginning of the main study through the end of the observational follow-up (up to 11.4 years)
Population: as for outcome 34
Measure: Number; unit: participants
Arm/Group | Combined RSG: Main Study and Observational Follow-up | Combined MET/SU: Main Study and Observational Follow-up
Number analyzed (Participants) | 2220 | 2227
participants
  Any cancer-related death | 59 | 72
  Any gastrointestinal event | 25 | 34
  Pancreatic | 4 | 12
  Colon/rectal | 6 | 11
  Gastric | 7 | 3
  Liver | 4 | 4
  Gall bladder/biliary | 4 | 3
  Gastrointestinal event; not specified | 0 | 1
  Any genitourinary event | 6 | 15
  Renal | 2 | 3
  Uterine | 1 | 5
  Prostate | 1 | 2
  Bladder | 1 | 3
  Ovarian | 1 | 2
  Lung | 13 | 11
  Any hematologic event | 4 | 0
  Skin (melanoma) | 3 | 0
  Skin (non-melanomatous) | 1 | 0
  Metastases | 2 | 4
  Breast | 2 | 3
  Head and neck | 1 | 2
  Any neurologic event | 2 | 2
  Endocrine | 1 | 0
  Not specified | 0 | 1

39. Secondary Outcome: Number of Participants Who Died Due to the Indicated Cancer-related Event: Observational Follow-up
Description: as for outcome 34
Time Frame: From the end of the RECORD study through the end of the observational follow-up (up to 4.0 years)
Population: as for outcome 35
Measure: Number; unit: participants
Arm/Group | Combined RSG: Observational Follow-up | Combined MET/SU: Observational Follow-up
Number analyzed (Participants) | 1280 | 1250
participants
  Any cancer-related death | 25 | 24
  Any gastrointestinal event | 10 | 14
  Pancreatic | 3 | 3
  Colon/rectal | 2 | 6
  Gastric | 2 | 1
  Liver | 2 | 2
  Gall bladder/biliary | 1 | 1
  Gastrointestinal event; not specified | 0 | 1
  Any genitourinary event | 2 | 0
  Renal | 1 | 0
  Uterine | 1 | 0
  Prostate | 0 | 0
  Bladder | 0 | 0
  Ovarian | 0 | 0
  Lung | 4 | 5
  Any hematologic event | 4 | 0
  Skin (melanoma) | 1 | 0
  Skin (non-melanomatous) | 1 | 0
  Metastases | 1 | 1
  Breast | 1 | 3
  Head and neck | 1 | 0
  Any neurologic event | 1 | 1
  Endocrine | 0 | 0
  Not specified | 0 | 0

40. Secondary Outcome: Number of Participants With a Bone Fracture Event - Overall and by Gender: Main Study and Observational Follow-up Combined
Description: The observational follow-up was designed to collect data concerning cancer and bone fractures in RECORD participants during a 4-year period after the end of the main RECORD study. At the end of the main study, all study medication was stopped. Participants were not provided with study medication in the observational follow-up; instead, anti-diabetic treatment was prescribed at the investigator's discretion. A bone fracture event is defined as one or more fractured bones occurring on the same date and that had the same Higher Level Group Term (HLGT) for fracture location, per participant.
Time Frame: From the beginning of the main study through the end of the observational follow-up (up to 11.4 years)
Population: as for outcome 34
Measure: Number; unit: participants
Arm/Group | Combined RSG: Main Study and Observational Follow-up | Combined MET/SU: Main Study and Observational Follow-up
Number analyzed (Participants) | 2220 | 2227
participants
  Overall, n=2220, 2227 | 238 | 151
  Male, n=1142, 1152 | 82 | 60
  Female, n=1078, 1075 | 156 | 91

41. Secondary Outcome: Number of Participants With a Bone Fracture Event - Overall and by Gender: Observational Follow-up
Description: as for outcome 40
Time Frame: From the end of the RECORD study through the end of the observational follow-up (up to 4.0 years)
Population: as for outcome 35
Measure: Number; unit: participants
Arm/Group | Combined RSG: Observational Follow-up | Combined MET/SU: Observational Follow-up
Number analyzed (Participants) | 1280 | 1250
participants
  Overall, n=1280, 1250 | 64 | 37
  Male, n=665, 635 | 25 | 11
  Female, n=615, 615 | 39 | 26

42. Secondary Outcome: Number of Participants With a Bone Fracture Event Reported as the Indicated Serious Adverse Event (by Higher Level Group Term) or Death: Main Study + Observational Follow-up Combined
Description: The OFU was designed to collect data concerning cancer and bone fractures in RECORD participants during a 4-year period after the end of the main RECORD study. At the end of the main study, all study medication was stopped. Participants were not provided with study medication in the OFU. A bone fracture event is defined as one or more fractured bones occurring on the same date and that had the same Higher Level Group Term (HLGT) for fracture location, per participant. An SAE is defined as any event that is fatal; life threatening; disabling/incapacitating; results in hospitalization (excluding elective surgery or routine clinical procedures); prolongs a hospital stay; is associated with a congenital abnormality; cancer; is associated with an overdose. In addition, any event that the investigator regards as serious or that would suggest any significant hazard, contraindication, side effect, or precaution that may be associated with the study procedures should be reported as an SAE.
Time Frame: From the beginning of the main study through the end of the observational follow-up (up to 11.4 years)
Population: as for outcome 34
Measure: Number; unit: participants
Arm/Group | Combined RSG: Main Study and Observational Follow-up | Combined MET/SU: Main Study and Observational Follow-up
Number analyzed (Participants) | 2220 | 2227
participants
  Any event | 81 | 57
  Upper limb | 41 | 17
  Distal lower limb | 24 | 16
  Femur/hip | 15 | 11
  Spinal | 7 | 9
  Pelvic | 0 | 3
  Other | 7 | 4

43. Secondary Outcome: Number of Participants With a Bone Fracture Event Reported as the Indicated Serious Adverse Event (by Higher Level Group Term) or Death: Observational Follow-up
Description: as for outcome 42
Time Frame: From the end of the RECORD study through the end of the observational follow-up (up to 4.0 years)
Population: as for outcome 35
Measure: Number; unit: participants
Arm/Group | Combined RSG: Observational Follow-up | Combined MET/SU: Observational Follow-up
Number analyzed (Participants) | 1280 | 1250
participants
  Any event | 35 | 21
  Upper limb | 17 | 5
  Distal lower limb | 9 | 8
  Femur/hip | 6 | 4
  Spinal | 2 | 3
  Pelvic | 0 | 1
  Other | 2 | 1

44. Secondary Outcome: Number of Participants With an Event of Death Due to a Bone Fracture-related Event: Main Study + Observational Follow-up Combined
Description: as for outcome 40
Time Frame: From the beginning of the main study through the end of the observational follow-up (up to 11.4 years)
Population: as for outcome 34
Measure: Number; unit: participants
Arm/Group | Combined RSG: Main Study and Observational Follow-up | Combined MET/SU: Main Study and Observational Follow-up
Number analyzed (Participants) | 2220 | 2227
participants | 0 | 0

45. Secondary Outcome: Number of Participants With the Indicated Bone Fracture by Fracture Site: Main Study + Observational Follow-up Combined
Description: The observational follow-up was designed to collect data concerning cancer and bone fractures in RECORD participants during a 4-year period after the end of the main RECORD study. At the end of the main study, all study medication was stopped. Participants were not provided with study medication in the observational follow-up; instead, anti-diabetic treatment was prescribed at the investigator's discretion. A bone fracture event is defined as one or more fractured bones occurring on the same date that had the same Higher Level Group Term (HLGT) for fracture location, per participant.
Time Frame: From the beginning of the main study through the end of the observational follow-up (up to 11.4 years)
Population: as for outcome 34
Measure: Number; unit: participants
Arm/Group | Combined RSG: Main Study and Observational Follow-up | Combined MET/SU: Main Study and Observational Follow-up
Number analyzed (Participants) | 2220 | 2227
participants
  Any event, overall; n=2220, 2227 | 238 | 151
  Any event, male; n=1142, 1152 | 82 | 60
  Any event, female; n=1078, 1075 | 156 | 91
  Upper limb, any event, overall; n=2220, 2227 | 116 | 70
  Upper limb, any event, male; n=1142, 1152 | 32 | 22
  Upper limb, any event, female; n=1078, 1075 | 84 | 48
  Distal lower limb, any event, overall; n=2220, 222 | 88 | 40
  Distal lower limb, any event, male; n=1142, 1152 | 31 | 14
  Distal lower limb, any event, female; n=1078, 1075 | 57 | 26
  Femur/hip, any event, overall; n=2220, 2227 | 16 | 13
  Femur/hip, any event, male; n=1142, 1152 | 4 | 1
  Femur/hip, any event, female; n=1078, 1075 | 12 | 12
  Spinal, any event, overall; n=2220, 2227 | 18 | 14
  Spinal, any event, male; n=1142, 1152 | 7 | 9
  Spinal, any event, female; n=1078, 1075 | 11 | 5
  Pelvic, any event, overall; n=2220, 2227 | 0 | 5
  Pelvic, any event, male; n=1142, 1152 | 0 | 4
  Pelvic, any event, female; n=1078, 1075 | 0 | 1
  Unclassified, any event, overall; n=2220, 2227 | 1 | 0
  Unclassified, any event, male; n=1142, 1152 | 1 | 0
  Unclassified, any event, female; n=1078, 1075 | 0 | 0
  Other, any event, overall; n=2220, 2227 | 31 | 26
  Other, any event, male; n=1142, 1152 | 18 | 16
  Other, any event, female; n=1078, 1075 | 13 | 10

46. Secondary Outcome: Number of Participants With the Indicated Bone Fracture by Fracture Site: Observational Follow-up
Description: as for outcome 45
Time Frame: From the end of the RECORD study through the end of the observational follow-up (up to 4.0 years)
Population: as for outcome 35
Measure: Number; unit: participants
Arm/Group | Combined RSG: Observational Follow-up | Combined MET/SU: Observational Follow-up
Number analyzed (Participants) | 1280 | 1250
participants
  Any event, overall; n=1280, 1250 | 64 | 37
  Any event, male; n=665, 635 | 25 | 11
  Any event, female; n=615, 615 | 39 | 26
  Upper limb, any event, overall; n=1280, 1250 | 33 | 15
  Upper limb, any event, male; n=665, 635 | 10 | 3
  Upper limb, any event, female; n=615, 615 | 23 | 12
  Distal lower limb, any event, overall; n=1280,1250 | 18 | 13
  Distal lower limb, any event, male; n=665, 635 | 9 | 4
  Distal lower limb, any event, female; n=615, 615 | 9 | 9
  Femur/hip, any event, overall; n=1280, 1250 | 6 | 5
  Femur/hip, any event, male; n=665, 635 | 1 | 0
  Femur/hip, any event, female; n=615, 615 | 5 | 5
  Spinal, any event, overall; n=1280, 1250 | 4 | 5
  Spinal, any event, male; n=665, 635 | 1 | 4
  Spinal, any event, female; n=615, 615 | 3 | 1
  Pelvic, any event, overall; n=1280, 1250 | 0 | 1
  Pelvic, any event, male; n=665, 635 | 0 | 1
  Pelvic, any event, female; n=615, 615 | 0 | 0
  Unclassified, any event, overall; n=1280, 1250 | 1 | 0
  Unclassified, any event, male; n=665, 635 | 1 | 0
  Unclassified, any event, female; n=615, 615 | 0 | 0
  Other, any event, overall; n=1280, 1250 | 6 | 1
  Other, any event, male; n=665, 635 | 4 | 1
  Other, any event, female; n=615, 615 | 2 | 0

47. Secondary Outcome: Number of Participants With Potentially High Morbidity Fractures: Main Study + Observational Follow-up Combined
Description: The observational follow-up was designed to collect data concerning cancer and bone fractures in RECORD participants during a 4-year period after the end of the main RECORD study. At the end of the main study, all study medication was stopped. Participants were not provided with study medication in the observational follow-up; instead, anti-diabetic treatment was prescribed at the investigator's discretion. A bone fracture event is defined as one or more fractured bones occurring on the same date and that had the same Higher Level Group Term (HLGT) for fracture location, per participant. The following bone fractures were grouped and were identified as potentially high morbidity bone fractures: hip, pelvis, upper leg, vertebral (lumbar spine, thoracic spine, cervical spine, spine - site unknown).
Time Frame: From the beginning of the main study through the end of the observational follow-up (up to 11.4 years)
Population: as for outcome 34
Measure: Number; unit: participants
Arm/Group | Combined RSG: Main Study and Observational Follow-up | Combined MET/SU: Main Study and Observational Follow-up
Number analyzed (Participants) | 2220 | 2227
participants
  Any event, overall, n=2220, 2227 | 31 | 31
  Any event, male, n=1142, 1152 | 10 | 13
  Any event, female, n=1078, 1075 | 21 | 18
  Hip, overall, n=2220, 2227 | 9 | 7
  Hip, male, n=1142, 1152 | 0 | 1
  Hip, female, n=1078, 1075 | 9 | 6
  Pelvis, overall, n=2220, 2227 | 0 | 5
  Pelvis, male, n=1142, 1152 | 0 | 4
  Pelvis, female, n=1078, 1075 | 0 | 1
  Upper leg, overall, n=2220, 2227 | 7 | 6
  Upper leg, male, n=1142, 1152 | 4 | 0
  Upper leg, female, n=1078, 1075 | 3 | 6
  Any vertebral event, overall, n=2220, 2227 | 16 | 13
  Any vertebral event, male, n=1142, 1152 | 6 | 8
  Any vertebral event, female, n=1078, 1075 | 10 | 5
  Lumbar spine, overall, n=2220, 2227 | 10 | 4
  Lumbar spine, male, n=1142, 1152 | 5 | 3
  Lumbar spine, female, n=1078, 1075 | 5 | 1
  Thoracic spine, overall, n=2220, 2227 | 5 | 8
  Thoracic spine, male, n=1142, 1152 | 1 | 4
  Thoracic spine, female, n=1078, 1075 | 4 | 4
  Cervical spine, overall, n=2220, 2227 | 1 | 1
  Cervical spine, male, n=1142, 1152 | 0 | 1
  Cervical spine, female, n=1078, 1075 | 1 | 0

48. Secondary Outcome: Number of Participants With Potentially High Morbidity Fracture Events and Non-high Morbidity Fracture Events, in Participants With Prior Hand/Upper Arm/Foot Fractures (H/UA/FF): Main Study + Observational Follow-up Combined
Description: as for outcome 47
Time Frame: From the beginning of the main study through the end of the observational follow-up (up to 11.4 years)
Population: as for outcome 34
Measure: Number; unit: participants
Arm/Group | Combined RSG: Main Study and Observational Follow-up | Combined MET/SU: Main Study and Observational Follow-up
Number analyzed (Participants) | 2220 | 2227
participants
  Any H/UA/FF event, overall, n=2220, 2227 | 86 | 46
  Any H/UA/FF event, male, n=1142, 1152 | 28 | 15
  Any H/UA/FF event, female, n=1078, 1075 | 58 | 31
  High morbidity fractures, overall, n=2220, 2227 | 5 | 1
  High morbidity fractures, male, n=1142, 1152 | 0 | 0
  High morbidity fractures, female, n=1078, 1075 | 5 | 1
  Non-high morbidity fractures, overall, n=2220, 222 | 15 | 4
  Non-high morbidity fractures, male, n=1142, 1152 | 2 | 3
  Non-high morbidity fractures, female, n=1078, 1075 | 13 | 1

49. Secondary Outcome: Number of Participants With Bone Fracture Events of the Indicated Cause: Main Study + Observational Follow-up Combined
Description: as for outcome 40
Time Frame: From the beginning of the main study through the end of the observational follow-up (up to 11.4 years)
Population: as for outcome 34
Measure: Number; unit: participants
Arm/Group | Combined RSG: Main Study and Observational Follow-up | Combined MET/SU: Main Study and Observational Follow-up
Number analyzed (Participants) | 2220 | 2227
participants
  Any event | 238 | 151
  Non-traumatic event | 113 | 55
  Traumatic event | 110 | 77
  Pathologic | 1 | 4
  Unknown | 20 | 19
  Data unavailable | 9 | 3

50. Secondary Outcome: Number of Participants With Bone Fracture Events of the Indicated Cause: Observational Follow-up
Description: The observational follow-up was designed to collect data concerning cancer and bone fractures in RECORD participants during a 4-year period after the end of the main RECORD study. At the end of the main study, all study medication was stopped. Participants were not provided with study medication in the observational follow-up; instead, anti-diabetic treatment was prescribed at the investigator's discretion. A bone fracture event is defined as one or more fractured bones occurring on the same date and that had the same Higher Level Group Term (HLGT) for fracture location, per participant. The indicated fracture outcome was pre-specified in the CRF and included "Unknown" as a category. Fracture events with missing outcome data were reported as "Data unavailable."
Time Frame: From the end of the RECORD study through the end of the observational follow-up (up to 4.0 years)
Population: as for outcome 35
Measure: Number; unit: participants
Arm/Group | Combined RSG: Observational Follow-up | Combined MET/SU: Observational Follow-up
Number analyzed (Participants) | 1280 | 1250
participants
  Any event | 64 | 37
  Non-traumatic event, | 36 | 14
  Traumatic event | 24 | 17
  Pathologic | 1 | 2
  Unknown | 1 | 4
  Data unavailable | 3 | 1

51. Secondary Outcome: Number of Bone Fracture Events With the Indicated Outcome: Main Study + Observational Follow-up Combined
Description: as for outcome 50
Time Frame: From the beginning of the main study through the end of the observational follow-up (up to 11.4 years)
Population: as for outcome 34
Measure: Number; unit: bone fracture events
Arm/Group | Combined RSG: Main Study and Observational Follow-up | Combined MET/SU: Main Study and Observational Follow-up
Number analyzed (Participants) | 2220 | 2227
bone fracture events
  Number of bone fracture events | 299 | 174
  Unknown | 7 | 5
  Normal healing with standard management | 250 | 142
  Complication | 14 | 13
  Additional therapeutic measures required | 16 | 9
  Data unavailable | 12 | 5

52. Secondary Outcome: Number of Bone Fracture Events With the Indicated Outcome: Observational Follow-up
Description: as for outcome 50
Time Frame: From the end of the RECORD study through the end of the observational follow-up (up to 4.0 years)
Population: as for outcome 35
Measure: Number; unit: bone fracture events
Arm/Group | Combined RSG: Observational Follow-up | Combined MET/SU: Observational Follow-up
Number analyzed (Participants) | 1280 | 1250
bone fracture events
  Number of bone fracture events | 70 | 41
  Unknown | 1 | 1
  Normal healing with standard management | 51 | 33
  Complication | 7 | 4
  Additional therapeutic measures required | 3 | 2
  Data unavailable | 8 | 1

53. Secondary Outcome: Number of Participants With the Indicated Serious Adverse Event: Observational Follow-up
Description: as for outcome 34
Time Frame: From the end of the RECORD study through the end of the observational follow-up (up to 4.0 years)
Population: as for outcome 35
Measure: Number; unit: participants
Arm/Group | Combined RSG: Observational Follow-up | Combined MET/SU: Observational Follow-up
Number analyzed (Participants) | 1280 | 1250
participants
  Any event | 99 | 76
  Ankle fracture | 6 | 3
  Prostate cancer | 7 | 1
  Lung neoplasm malignant | 4 | 4
  Breast cancer | 2 | 6
  Basal cell carcinoma | 4 | 3
  Pancreatic carcinoma | 4 | 3
  Colon cancer | 1 | 6
  Humerus fracture | 5 | 1
  Upper limb fracture | 5 | 1
  Malignant melanoma | 3 | 2
  Uterine cancer | 2 | 3
  Gastric cancer | 4 | 0
  Wrist fracture | 4 | 0
  Hip fracture | 3 | 1
  Radius fracture | 3 | 1
  Forearm fracture | 2 | 2
  Hepatic neoplasm malignant | 2 | 2
  Rectal cancer | 2 | 2
  Renal cancer | 2 | 2
  Foot fracture | 1 | 3
  Renal cell carcinoma | 3 | 0
  Femur fracture | 2 | 1
  Femoral neck fracture | 1 | 2
  Lumbar vertebral fracture | 1 | 2
  Metastases to bone | 1 | 2
  Metastases to liver | 1 | 2
  Bladder cancer | 2 | 0
  Fall | 2 | 0
  Metastases to central nervous system | 2 | 0
  Rib fracture | 2 | 0
  Squamous cell carcinoma | 2 | 0
  Acute myocardial infarction | 1 | 1
  Brain neoplasm | 1 | 1
  Gastric neoplasm | 1 | 1
  Metastases to lung | 1 | 1
  Patella fracture | 1 | 1
  Death | 0 | 2
  Abdominal pain | 1 | 0
  Acute myeloid leukaemia | 1 | 0
  Acute respiratory failure | 1 | 0
  Anaemia | 1 | 0
  Benign salivary gland neoplasm | 1 | 0
  Biliary colic | 1 | 0
  Biliary neoplasm | 1 | 0
  Bone neoplasm malignant | 1 | 0
  Bronchial carcinoma | 1 | 0
  Cardiac failure acute | 1 | 0
  Chest pain | 1 | 0
  Chronic lymphocytic leukaemia | 1 | 0
  Colon neoplasm | 1 | 0
  Contusion | 1 | 0
  Drowning | 1 | 0
  Dysplasia | 1 | 0
  Endometrial cancer stage I | 1 | 0
  Leukaemia | 1 | 0
  Lower limb fracture | 1 | 0
  Lung squamous cell carcinoma stage unspecified | 1 | 0
  Lymphoma | 1 | 0
  Malignant neoplasm of pleura | 1 | 0
  Metastases to skin | 1 | 0
  Metastases to testicle | 1 | 0
  Metastatic renal cell carcinoma | 1 | 0
  Oesophageal carcinoma | 1 | 0
  Osteoarthritis | 1 | 0
  Pancreatic necrosis | 1 | 0
  Rectal cancer stage II | 1 | 0
  Spinal fracture | 1 | 1
  T-cell lymphoma | 1 | 1
  Urinary tract infection | 1 | 1
  Uterine leiomyosarcoma | 1 | 0
  Biliary cancer metastatic | 0 | 1
  Cervix carcinoma | 0 | 1
  Chronic obstructive pulmonary disease | 0 | 1
  Comminuted fracture | 0 | 1
  Craniocerebral injury | 0 | 1
  Gastrointestinal neoplasm | 0 | 1
  Hepatic lesion | 0 | 1
  Joint dislocation | 0 | 1
  Laryngeal cancer | 0 | 1
  Lip neoplasm malignant stage unspecified | 0 | 1
  Lung neoplasm | 0 | 1
  Metastases to lymph nodes | 0 | 1
  Metastasis | 0 | 1
  Musculoskeletal chest pain | 0 | 1
  Myocardial infarction | 0 | 1
  Non-Hodgkin's lymphoma | 0 | 1
  Pubis fracture | 0 | 1
  Pulmonary embolism | 0 | 1
  Rectal cancer recurrent | 0 | 1
  Rectal neoplasm | 0 | 1
  Skin cancer | 0 | 1
  Skin ulcer | 0 | 1
  Small cell lung cancer stage unspecified | 0 | 1
  Sternal fracture | 0 | 1
  Subdural haemorrhage | 0 | 1
  Sudden death | 0 | 1
  Thoracic vertebral fracture | 0 | 1
  Thyroid cancer | 0 | 1
  Vulval cancer | 0 | 1

ADVERSE EVENTS:
Time Frame: In the RECORD study (RS), SAEs were collected from BL through End of Study (up to 7.5 years); non-serious AEs were collected only for the randomized treatment period. SAEs were collected from the end of the RS through the end of OFU (up to 4.0 years).
Description: The Observational Follow-up was designed to collect data concerning cancer and bone fractures in RECORD participants during a 4-year period after the end of the main RECORD study. Other than bone fractures (tabulated in the Outcome Measure Module), no non-serious AEs were collected.
Arm/Group | RSG in Addition to Background MET | SU in Addition to Background MET | RSG in Addition to Background SU | MET in Addition to Background SU | Combined RSG: Observational Follow-up | Combined MET/SU: Observational Follow-up
Serious Adverse Events (participants affected / at risk) | 424/1117 | 428/1105 | 427/1103 | 431/1122 | 99/1280 | 76/1250
Other Adverse Events (participants affected / at risk) | 1117/1117 | 1105/1105 | 1103/1103 | 1122/1122 | 0/1280 | 0/1250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | RSG in Addition to Background MET (N=1117) | SU in Addition to Background MET (N=1105) | RSG in Addition to Background SU (N=1103) | MET in Addition to Background SU (N=1122) | Combined RSG: Observational Follow-up (N=1280) | Combined MET/SU: Observational Follow-up (N=1250)
Myocardial Infarction (Cardiac disorders) | 25 | 22 | 29 | 23 | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 25 | 18 | 23 | 13 | 0 | 0
Angina Pectoris (Cardiac disorders) | 23 | 18 | 23 | 19 | 0 | 0
Angina Unstable (Cardiac disorders) | 16 | 20 | 21 | 18 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 20 | 15 | 13 | 14 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 12 | 6 | 11 | 19 | 1 | 1
Cardiac Failure (Cardiac disorders) | 16 | 1 | 13 | 8 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 9 | 6 | 7 | 12 | 0 | 0
Myocardial Ischaemia (Cardiac disorders) | 7 | 5 | 7 | 5 | 0 | 0
Coronary Artery Stenosis (Cardiac disorders) | 4 | 8 | 5 | 7 | 0 | 0
Cardiac Failure Acute (Cardiac disorders) | 3 | 2 | 3 | 3 | 1 | 0
Arrythmia (Cardiac disorders) | 1 | 4 | 2 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 3 | 1 | 0 | 0 | 0
Acute Coronary Syndrome (Cardiac disorders) | 3 | 0 | 0 | 1 | 0 | 0
Arteriosclerosis Coronary Artery (Cardiac disorders) | 2 | 1 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 1 | 0 | 0 | 0 | 0
Atrioventricular Block Complete (Cardiac disorders) | 1 | 2 | 0 | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 2 | 0 | 0 | 0 | 0
Aortic Valve Disease (Cardiac disorders) | 2 | 0 | 0 | 1 | 0 | 0
Sick Sinus Syndrome (Cardiac disorders) | 2 | 0 | 1 | 0 | 0 | 0
Atrial Flutter (Cardiac disorders) | 1 | 1 | 1 | 4 | 0 | 0
Cardiac Disorder (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0
Silent Myocardial Infarction (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0
Mitral Valve Incompetence (Cardiac disorders) | 0 | 2 | 0 | 1 | 0 | 0
Atrial Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrioventricular Block Second Degree (Cardiac disorders) | 1 | 0 | 2 | 0 | 0 | 0
Cardiac Failure Chronic (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cor pulmonale (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Left Ventricular Failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mitral Valve Disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0
Right Ventricular Failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 2 | 0 | 0
Ventricular Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ventricular Fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Congestive Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 2 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 1 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1 | 2 | 0 | 0
Aortic Valve Stenosis (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0
Coronary Artery Occlusion (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Tachycardia Paroxysmal (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Atrioventricular Block (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0
Bradyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0
Cardiac Fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cardiac Flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Adams-Stokes Syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertensive Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Left Ventricular Hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myocardial Fibrosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Supraventricular Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tricuspid Valve Incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pnuemonia (Infections and infestations) | 21 | 15 | 11 | 12 | 0 | 0
Erysipelas (Infections and infestations) | 6 | 7 | 6 | 1 | 0 | 0
Sepsis (Infections and infestations) | 6 | 5 | 4 | 3 | 0 | 0
Cellulitis (Infections and infestations) | 4 | 6 | 3 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 6 | 4 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 6 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 4 | 2 | 3 | 5 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 2 | 4 | 0 | 0 | 0 | 0
Bronchopnuemonia (Infections and infestations) | 1 | 5 | 4 | 1 | 0 | 0
Gangrene (Infections and infestations) | 0 | 4 | 3 | 4 | 0 | 0
Diverticulitis (Infections and infestations) | 2 | 1 | 2 | 5 | 0 | 0
Abdominal Abscess (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 2 | 2 | 5 | 0 | 0
Post Procedural Infection (Infections and infestations) | 1 | 2 | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0
Localised Infection (Infections and infestations) | 0 | 3 | 0 | 1 | 0 | 0
Postoperative Wound Infection (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0
Anal Abscess (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0
Orchitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Pyelonephritis Acute (Infections and infestations) | 0 | 2 | 3 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Abscess Intestinal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Appendiceal Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Bacterial Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Brochiectasis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Campylobacter Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis Infective (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Encephalitis Viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Endocarditis Viral (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Herpes Zoster (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Infective Exacercbatn of Chronic Obstructive Airways Disease (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Infective Thrombosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Joint Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Liver Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Mastitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Myocardiac Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 2 | 1 | 0 | 0
Pelvic Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Phlebitis Infective (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Retroperitoneal Abscess (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Toxoplasmosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Viral Infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Wound Infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 4 | 2 | 0 | 0
Arthritis Bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Catheter Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis Viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0
Enteritis Infectious (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis Bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Groin Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Hepatitis C (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Herpes Zoster Oticus (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Infective Myositis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Intestinal Gangrene (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Lobar Pneumonia (Infections and infestations) | 0 | 1 | 4 | 0 | 0 | 0
Lung Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Lyme Disease (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Meningitis Viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Necrotising Fasciitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Otitis Media Acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pancreatic Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Peridiverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Periumbilical Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumococcal Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia Bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Post Procedural Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pyelonephritis Chronic (Infections and infestations) | 0 | 1 | 1 | 2 | 0 | 0
Scrotal Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sialoadenitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Staphylococcal Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 3 | 1 | 0 | 0
Pulmonary Tuberculosis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Abdominal Wall Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Device Related Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Escherichia Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Extradural Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Hepatitis Viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Infected Cyst (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia Legionella (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pyelocystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urethritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Arteriosclerotic Gangrene (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Blister Infected (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Carbuncle (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Colostomy Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Diabetic Gangrene (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Ear Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis Salmonella (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Herpes Ophthalmic (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Keratitis herpetic (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Peritoneal Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pyothorax (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 9 | 5 | 8 | 7 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 4 | 4 | 3 | 4 | 3
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5 | 3 | 6 | 1 | 6
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3 | 1 | 3 | 2 | 6
Breast Cancer Female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 3 | 4 | 0 | 0
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5 | 3 | 0 | 2 | 2
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 6 | 1 | 5 | 4 | 3
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 1 | 4 | 1 | 2
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5 | 6 | 1 | 4 | 4
Gallbladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0 | 2 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 1 | 2 | 2 | 2
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 3 | 0 | 2 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 5 | 1 | 4 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 2 | 0 | 3 | 2
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 1 | 1 | 0
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 3 | 3 | 2 | 3
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2 | 2 | 0 | 0
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 3 | 0 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 2 | 2 | 0
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1 | 2 | 2
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0
Ovarian Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 1 | 3 | 0
Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 3 | 3 | 0 | 0
Prostatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 2 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Benign Salivary Gland Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 1 | 1 | 0
Gastrointestinal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Hairy Cell Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 1 | 0
Metastases to Abdominal Cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0
Nasal Cavity Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Ovarian Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0
Thyroid Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Wall Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Adrenocortical Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Bladder Transitional Cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 1 | 1
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0
Breast Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1 | 1 | 0
Colon Cancer Stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 1 | 0 | 0
Epiglottic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Metastases to Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1 | 1 | 1
Metastases to Lymph Nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Myeloproliferative Disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Oesophageal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 3 | 1 | 0 | 0
Ovarian Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Pancreatic Carcinoma Stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Rectal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0
Renal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Uterine Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 1 | 0
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 1 | 2 | 0
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1 | 0 | 0
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0
Rectal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 1
Benign Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Lip Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Metastases to Peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Metastatic Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Neoplasm Prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Pharyngeal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Vulval Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Hair Follicle Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Hepatic Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Malignant Mesenchymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Metastases to Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 2
Metastases to Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Metastases to Spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Metastatic Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Ovarian Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Rectal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Testicular Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Tongue Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 18 | 25 | 21 | 24 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 11 | 14 | 11 | 11 | 0 | 0
Syncope (Nervous system disorders) | 5 | 2 | 3 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 3 | 2 | 2 | 3 | 0 | 0
Carotid Artery Stenosis (Nervous system disorders) | 1 | 4 | 1 | 3 | 0 | 0
Diabetic Neuropathy (Nervous system disorders) | 3 | 1 | 3 | 2 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 3 | 1 | 2 | 7 | 0 | 0
Epilepsy (Nervous system disorders) | 3 | 0 | 0 | 2 | 0 | 0
Syncope Vasovagal (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0
Carpal Tunnel syndrome (Nervous system disorders) | 1 | 2 | 2 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 3 | 0 | 0 | 0 | 0
Cerebral Haemorrhage (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0
Dementia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Facial Paresis (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0
Global Amnesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 1 | 1 | 2 | 0 | 0
Loss of Consciousness (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 2 | 1 | 3 | 0 | 0
Cognitive Disorder (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0
Vertebrobasilar Insufficiency (Nervous system disorders) | 0 | 2 | 4 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhage Intracranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hemiplegia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Intracranial Haematoma (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Multiple Sclerosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Radiculopathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Vascular Dementia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vascular Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 2 | 0 | 0
Demyelination (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhagic Stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoxic Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ischaemic Cerebral Infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Normal Pressure Hydrocephalus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Paralysis (Nervous system disorders) | 0 | 1 | 0 | 2 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Reversible Ischaemic Neurological Deficit (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ruptured Cerebral Aneurysm (Nervous system disorders) | 0 | 1 | 0 | 0/1112 | 0 | 0
Tension Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cerebral Ischaemia (Nervous system disorders) | 0 | 0 | 4 | 2/1112 | 0 | 0
Brain Oedema (Nervous system disorders) | 0 | 0 | 1 | 0/1112 | 0 | 0
Cerebrovascular Insufficiency (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cervicobrachial Syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypertonia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Radiculitis lumbosacral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Carotid Arteriosclerosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cerebral Arteriosclerosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular Disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Facial Palsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertensive Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypokinesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lumbar Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Metabolic Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nerve Compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nerve Root Compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Parkinsonism (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 5 | 5 | 0 | 1 | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 6 | 3 | 4 | 1 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3 | 3 | 2 | 3 | 0 | 0
Gastritis (Gastrointestinal disorders) | 3 | 2 | 3 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 2 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0 | 0
Duodenal ulcer Haemorrhage (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 0 | 0
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 0
Umbilical Hernia (Gastrointestinal disorders) | 2 | 1 | 0 | 3 | 0 | 0
Crohn's Disease (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0
Gastric Polyps (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hiatus Hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 3 | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 0 | 0
Intestinal Perforation (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Abdominal Hernia Obstructive (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diverticulum Intestinal (Gastrointestinal disorders) | 1 | 0 | 1 | 4 | 0 | 0
Faeces Discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastric Dysplasia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 0 | 0
Gastritis Haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal Inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intestinal Fistula (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pancreatic Pseudocyst (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Peritoneal Disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Splenic Artery Aneurysm (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 0 | 0
Abdominal Hernia (Gastrointestinal disorders) | 0 | 1 | 2 | 2 | 0 | 0
Anal Fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Appendicitis Perforated (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Colonic Fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Colonic Polyp (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 0 | 0
Diverticular Perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diverticulitis Intestinal Haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Duodenal Perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Mechanical Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Reflux Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Small Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis Chronic (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0
Gastric Ulcer Perforation (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Abdominal Adhesions (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Gastroduodenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Pancreatic Cyst (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Pancreatitis Necrotising (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Peptic Ulcer Perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Duodenal Fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastroduodenal Ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pancreatic necrosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rectal Polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Salivary Gland Calculus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Duodenitis Haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Enterocele (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Intestinal Polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peptic Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 4 | 2 | 2 | 2 | 6 | 3
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 5 | 4 | 3 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 5 | 0 | 1 | 3 | 5 | 1
Fall (Injury, poisoning and procedural complications) | 4 | 1 | 3 | 1 | 2 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 3 | 2 | 3 | 0 | 3 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 1 | 2 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 3 | 1 | 2 | 4 | 5 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 2 | 2 | 2 | 1 | 3 | 1
Post Procedural Complication (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 1 | 0 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 0 | 0
Head Injury (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 2 | 0 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 1 | 0 | 1
Meniscus Lesion (Injury, poisoning and procedural complications) | 1 | 2 | 5 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 2 | 0 | 0
Drug Toxicity (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0
Facial Bones Fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0
Incisional Hernia (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0 | 0
Joint Injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0
Post Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 1 | 3 | 0 | 0 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0
Device Failure (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 1 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 2 | 0
Alcohol Poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac Valve Replacement Complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Cartilage Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0
Dislocation of Joint Prosthesis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Gun Shot Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1 | 2
Lung Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Multiple Fractures (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0
Near Drowning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Post Procedural Fistula (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Postoperative Ileus (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Skull Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Accident (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2 | 0 | 0
Acetabulum Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Anastomotic Leak (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 5 | 0 | 2 | 1
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 0 | 0
In-Stent Arterial Restenosis (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0
Multiple Injuries (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0 | 0 | 0
Muscle Rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 0 | 0
Stent Occlusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 1 | 3
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 1 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0
Brain Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0
Arthropod Sting (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Asbestosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Epiphyseal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Eyeball Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Intentional Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Joint Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Open Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Shunt Occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Synovial Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 4 | 0
Fibula Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Limb Crushing Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Limb Traumatic Amputation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Operative Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 1
Post Laminectomy Syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Post-Traumatic Pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Postoperative Hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Traumatic Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 7 | 10 | 10 | 10 | 0 | 0
Thrombosis (Vascular disorders) | 3 | 2 | 1 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 2 | 3 | 3 | 1 | 0 | 0
Aortic Stenosis (Vascular disorders) | 3 | 1 | 2 | 1 | 0 | 0
Intermittent Claudication (Vascular disorders) | 1 | 3 | 1 | 0 | 0 | 0
Varicose Vein (Vascular disorders) | 0 | 4 | 2 | 1 | 0 | 0
Aortic Aneurysm (Vascular disorders) | 2 | 0 | 1 | 0 | 0 | 0
Essential Hypertension (Vascular disorders) | 2 | 0 | 1 | 2 | 0 | 0
Hypovolaemic Shock (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 2 | 0 | 1 | 0 | 0 | 0
Femoral Artery Occlusion (Vascular disorders) | 1 | 1 | 1 | 3 | 0 | 0
Hypertensive Crisis (Vascular disorders) | 1 | 1 | 2 | 4 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 2 | 0 | 0
Shock (Vascular disorders) | 1 | 1 | 0 | 1 | 0 | 0
Iliac Artery Stenosis (Vascular disorders) | 0 | 2 | 1 | 0 | 0 | 0
Peripheral Ischaemia (Vascular disorders) | 0 | 2 | 2 | 3 | 0 | 0
Accelerated Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arteriosclerosis obliterans (Vascular disorders) | 1 | 0 | 1 | 1 | 0 | 0
Artery Dissection (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Circulatory Collapse (Vascular disorders) | 1 | 0 | 2 | 2 | 0 | 0
Diabetic Microangiopathy (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0
Shock Haemorrhagic (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Aortic Aneurysm Rupture (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arterial Occlusive Disease (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arterial Stenosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arterial Stenosis Limb (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cardiovascular Insufficiency (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0
Extremity Necrosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Femoral Arterial Stenosis (Vascular disorders) | 0 | 1 | 1 | 2 | 0 | 0
Labile Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Malignant Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 | 1 | 3 | 0 | 0 | 0
Peripheral Vascular Disorder (Vascular disorders) | 0 | 1 | 5 | 0 | 0 | 0
Thrombophlebitis Superficial (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0
Venous Insufficiency (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Venous Thrombosis Limb (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 5 | 0 | 0
Arterial Thrombosis Limb (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0
Angiopathy (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arterial Disorder (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ischaemia (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Venous Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diabetic Microangiopathy (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 16 | 12 | 13 | 12 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 3 | 4 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 2 | 5 | 6 | 6 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 3 | 0 | 0 | 0
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1 | 0 | 0
Dupuytren's Contracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 0 | 0
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 0 | 1
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | 5 | 0 | 0
Diabetic Amyotrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Senile Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rheumatic Fever (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 4 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Compartment Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 9 | 4 | 4 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 8 | 4 | 0 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0 | 4 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 1 | 0 | 0
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 0
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2 | 0 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0 | 0
Alveolitis Fibrosing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0 | 0
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 0 | 0
Lung Consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nasal Turbinate Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tracheal Stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysnoea Paroxysmal Nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nocturnal Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Respiratory Alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 14 | 12 | 5 | 3 | 0 | 0
Death (General disorders) | 5 | 3 | 2 | 6 | 0 | 2
Pyrexia (General disorders) | 4 | 2 | 3 | 0 | 0 | 0
Sudden Death (General disorders) | 1 | 3 | 4 | 4 | 0 | 1
Inflammation (General disorders) | 2 | 0 | 2 | 0 | 0 | 0
Multi-Organ Failure (General disorders) | 1 | 1 | 1 | 0 | 0 | 0
Sudden Cardiac Death (General disorders) | 1 | 1 | 2 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 2 | 0 | 0 | 1 | 0
Gait Disturbance (General disorders) | 0 | 2 | 0 | 0 | 0 | 0
Hernia Obstructive (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chest Discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
General Physical Health Deterioration (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Drowning (General disorders) | 0 | 0 | 0 | 2 | 1 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tenderness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Brain Death (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 15 | 13 | 9 | 10 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 5 | 5 | 4 | 3 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 2 | 2 | 5 | 1 | 0 | 0
Liver Disorder (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Biliary Colic (Hepatobiliary disorders) | 1 | 0 | 2 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hepatic Failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bile Duct Obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bile Duct Stone (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 0
Hepatic Steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Jaundice Cholestatic (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0 | 0
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0 | 0
Gallbladder Polyp (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatitis Alcoholic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Post Cholecystectomy Syndrome (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 5 | 10 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 9 | 6 | 9 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 4 | 5 | 10 | 17 | 0 | 0
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 2 | 3 | 2 | 10 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 0 | 0
Diabetic Foot (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemochromatosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Diabetic Complication (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypeonatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Podagra (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Increased Insulin Requirement (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 3 | 8 | 2 | 5 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 3 | 8 | 2 | 5 | 0 | 0
Renal Failure (Renal and urinary disorders) | 3 | 4 | 0 | 0 | 0 | 0
Renal Colic (Renal and urinary disorders) | 2 | 2 | 1 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 2 | 1 | 2 | 0 | 0 | 0
Calculus Ureteric (Renal and urinary disorders) | 1 | 2 | 1 | 1 | 0 | 0
Calculus Urinary (Renal and urinary disorders) | 1 | 2 | 2 | 3 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 2 | 1 | 0 | 0 | 0
Cystitis Noninfective (Renal and urinary disorders) | 0 | 2 | 0 | 1 | 0 | 0
Acute Prerenal Failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Urethral Fistula (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urinary Bladder Haemorrhage (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bladder Perforation (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diabetic Nephropathy (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urethral Stenosis (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0
Renal Cyst (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0
Albuminuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Calculus Bladder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Renal Pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary Tract Inflammation (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Calculus Urethral (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ketonuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal Embolism (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urine Flow Decreased (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 3 | 6 | 6 | 4 | 0 | 0
Uterine Prolapse (Reproductive system and breast disorders) | 0 | 4 | 0 | 2 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 2 | 0 | 0 | 1 | 0 | 0
Rectocele (Reproductive system and breast disorders) | 2 | 0 | 0 | 1 | 0 | 0
Breast Disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cervical Polyp (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Endometrial Hypertrophy (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0 | 0
Peyronie's Disease (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Testicular Pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vaginal Prolapse (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0 | 0
Fibrocystic Breast Disease (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0 | 0
Vaginal Cyst (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0 | 0
Vulvovaginal Dryness (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 0 | 0 | 2 | 1 | 0 | 0
Uterine Polyp (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0 | 0
Orchitis Noninfective (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pelvic Peritoneal Adhesions (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Prostatic Obstruction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Prostatism (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vaginal Polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vulval Leukoplakia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 5 | 3 | 12 | 9 | 0 | 0
Retinal Detachment (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0
Angle Closure Glaucoma (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0
Maculopathy (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 1 | 0 | 1 | 2 | 0 | 0
Cataract Nuclear (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Inflammation of Lacrimal Passage (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Retinal Haemorrhage (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0
Vitreous Haemorrhage (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0
Diabetic Retinopathy (Eye disorders) | 0 | 0 | 1 | 3 | 0 | 0
Eye Haemorrhage (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0
Dacryostenosis Acquired (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Exudative Retinopathy (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Macular Degeneration (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Optic Atrophy (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lens Dislocation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Retinal Vein Thrombosis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 8 | 2 | 4 | 5 | 1 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 2 | 0 | 0 | 0
Hypocoagulable State (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Idiopathic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Autoimmune Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 2 | 4 | 1 | 2 | 0 | 0
Confusional State (Psychiatric disorders) | 3 | 0 | 1 | 1 | 0 | 0
Alcohol Abuse (Psychiatric disorders) | 2 | 0 | 0 | 1 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 1 | 1 | 0 | 1 | 0 | 0
Mania (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bipolar Disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Completed Suicide (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysthymic Disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 4 | 6 | 5 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 2 | 0 | 0 | 1 | 0 | 0
Otosclerosis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sudden Hearing Loss (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1 | 2 | 0 | 0
Vestibular Disorder (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vestibular Neuronitis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vertigo Positional (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 2 | 2 | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 1 | 2 | 1 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperparathyroidism Primary (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Parathyroid Gland Enlargement (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Toxic Nodular Goitre (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Adrenal Mass (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0
Basedow's Disease (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 0 | 0 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lichen Planus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pityriasis Rubra Pilaris (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Blood glucose Increased (Investigations) | 1 | 1 | 2 | 4 | 0 | 0
Electrocardiogram T Wave Abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood Pressure Increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Liver Function Test Abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Weight Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood Urea Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Haemoglobin Decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Chest X-ray Abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 3 | 0 | 0 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Corneal Dystrophy (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 1 | 0 | 0
Gastrointestinal Angiodysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Splenic abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Malignant neoplasm of pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Metastases to testicle (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Rectal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Biliary cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Rectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 2
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Dysplasia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hepatic lesion (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RSG in Addition to Background MET (N=1117) | SU in Addition to Background MET (N=1105) | RSG in Addition to Background SU (N=1103) | MET in Addition to Background SU (N=1122) | Combined RSG: Observational Follow-up (N=1280) | Combined MET/SU: Observational Follow-up (N=1250)
Hypertension (Vascular disorders) | 345 | 372 | 302 | 319 | 0 | 0
Nasopharyngitis (Infections and infestations) | 216 | 202 | 121 | 122 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 236 | 144 | 193 | 120 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 153 | 143 | 95 | 105 | 0 | 0
Bronchitis (Infections and infestations) | 139 | 128 | 136 | 122 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 119 | 126 | 98 | 70 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 51 | 190 | 162 | 144 | 0 | 0
Influenza (Infections and infestations) | 110 | 129 | 106 | 88 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 121 | 78 | 155 | 64 | 0 | 0
Oedema peripheral (General disorders) | 144 | 47 | 133 | 41 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 60 | 81 | 44 | 135 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 81 | 79 | 61 | 51 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 105 | 45 | 55 | 38 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 51 | 97 | 49 | 68 | 0 | 0
Urinary tract infection (Infections and infestations) | 66 | 66 | 59 | 49 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 73 | 55 | 34 | 35 | 0 | 0
Headache (Nervous system disorders) | 66 | 61 | 58 | 47 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 59 | 67 | 54 | 42 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 73 | 45 | 81 | 57 | 0 | 0
Cataract (Eye disorders) | 51 | 66 | 56 | 67 | 0 | 0
Depression (Psychiatric disorders) | 67 | 47 | 34 | 35 | 0 | 0
Dizziness (Nervous system disorders) | 60 | 38 | 46 | 42 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 54 | 53 | 87 | 63 | 0 | 0
Diabetic retinopathy (Eye disorders) | 44 | 53 | 51 | 61 | 0 | 0
Viral infection (Infections and infestations) | 54 | 45 | 56 | 40 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 102 | 82 | 62 | 50 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.